CLINICAL TRIAL: NCT01402986
Title: A Phase 2b, Randomized, Double-blind Study to Evaluate the Efficacy of Tralokinumab in Adults With Uncontrolled, Severe Asthma
Brief Title: A Safety and Efficacy Study of Tralokinumab in Adults With Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CD-RI-CAT-354-1049; 2011-001360-21 (EudraCT Number)
Record Dates: First submitted 2011-07-21; First posted 2011-07-27 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Asthma
Keywords: Asthma; Tralokinumab; CAT-354
MeSH Terms: conditions — Asthma | interventions — tralokinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo, Q2W - Cohort 1 (Placebo Comparator): Participants received matching placebo subcutaneous injection every 2 weeks (Q2W) for a total of 26 doses up to 50 weeks.
  Interventions: Other: Placebo Q2W
- Tralokinumab 300 mg, Q2W - Cohort 1 (Experimental): Participants received tralokinumab 300 milligram (mg) subcutaneous injection every 2 weeks (Q2W) for a total of 26 doses up to 50 weeks.
  Interventions: Biological: Tralokinumab 300 mg, Q2W
- Placebo, Q2/4W - Cohort 2 (Placebo Comparator): Participants received matching placebo subcutaneous injection every 2 weeks (Q2W) for 12 weeks followed by every 4 weeks (Q4W) for 38 weeks (Q2/4W) for a total of 16 doses.
  Interventions: Other: Placebo, Q2/4W
- Tralokinumab 300 mg, Q2/4W - Cohort 2 (Experimental): Participants received tralokinumab 300 mg subcutaneous injection every 2 weeks (Q2W) for 12 weeks followed by every 4 weeks (Q4W) for 38 weeks (Q2/4W) for a total of 16 doses.
  Interventions: Biological: Tralokinumab 300 mg, Q2/4W

INTERVENTIONS:
Other: Placebo Q2W — Participants who received matching placebo subcutaneous injection every 2 weeks (Q2W) for a total of 26 doses up to 50 weeks.
  Arms: Placebo, Q2W - Cohort 1
Biological: Tralokinumab 300 mg, Q2W — Participants received tralokinumab 300 mg subcutaneous injection Q2W for a total of 26 doses up to 50 weeks.
  Other Names: CAT-354
  Arms: Tralokinumab 300 mg, Q2W - Cohort 1
Other: Placebo, Q2/4W — Participants received matching placebo subcutaneous injection Q2W for 12 weeks followed by Q4W for 38 weeks (Q2/4W) for a total of 16 doses.
  Arms: Placebo, Q2/4W - Cohort 2
Biological: Tralokinumab 300 mg, Q2/4W — Participants received tralokinumab 300 mg subcutaneous injection Q2W for 12 weeks followed by Q4W for 38 weeks (Q2/4W) for a total of 16 doses.
  Other Names: CAT-354
  Arms: Tralokinumab 300 mg, Q2/4W - Cohort 2

SUMMARY:
The purpose of this study is to determine whether the addition of tralokinumab to standard asthma medication is effective in the treatment of adults with asthma.

DETAILED DESCRIPTION:
Interleukin-13 (IL-13) is a key mediator in the pathogenesis of established asthmatic disease. Tralokinumab is a human monoclonal antibody that blocks IL-13, which may result in improved control of asthma. This study will determine whether the addition of tralokinumab to standard asthma medications results in a reduced rate of asthma exacerbations in subjects with severe asthma.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Body mass index (BMI) between 16-40 kilogram per square meter (kg/m^2) at Visit 1
* Uncontrolled severe asthma
* A chest x-ray with no abnormality
* Females of childbearing potential who are sexually active with a non-sterilized male partner must use highly effective contraception from Day 1
* Non-sterilized males or sterilized males who are less than or equal to (=<) 1 year post-vasectomy who are sexually active with a female partner of childbearing potential must use a highly effective method of contraception

Exclusion Criteria:

* Employee of the clinical study site or any other individuals directly involved with the conduct of the study, or immediate family members of such individuals
* Pregnant or breastfeeding women
* Any other respiratory disease
* Previously taken tralokinumab (the study drug)
* Current smoker or a history of smoking which would be more than 1 pack per day for 10 years
* Known immune deficiency
* History of cancer
* Hepatitis B, C or Human Immuno-deficiency Virus (HIV)
* Any disease which may cause complications whilst taking the study drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 689 (Actual)
Dates: Start 2011-08; Primary Completion 2013-06 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Piper, MBBS, Study Director — Sponsor GmbH; Christopher Brightling, Principal Investigator — Institute for Lung Health
Locations (89):
- United States (11):
  - Research Site, Rancho Mirage, California
  - Research Site, Centennial, Colorado
  - Research Site, New Haven, Connecticut
  - Research Site, Cocoa, Florida
  - Research Site, Miami, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Albany, Georgia
  - Research Site, Fargo, North Dakota
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Upland, Pennsylvania
  - Research Site, Killeen, Texas
- Argentina (5):
  - Research Site, Buenos Aires
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Monte Grande
  - Research Site, Ranelagh
  - Research Site, Rosario
- Canada (4):
  - Research Site, Calgary, Alberta
  - Research Site, Ottawa, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- Chile (4):
  - Research Site, Quillota
  - Research Site, Santiago
  - Research Site, Valparaíso
  - Research Site, Viña del Mar
- Czechia (3):
  - Research Site, Jindřichův Hradec
  - Research Site, Pilsen
  - Research Site, Rokycany
- France (7):
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Perpignan
  - Research Site, Pessac
  - Research Site, Strasbourg
- Germany (4):
  - Research Site, Berlin
  - Research Site, Frankfurt
  - Research Site, Lübeck
  - Research Site, Mainz
- Japan (22):
  - Research Site, Chūōku
  - Research Site, Fujisawa-shi
  - Research Site, Fukuoka
  - Research Site, Habikino-shi
  - Research Site, Hiroshima
  - Research Site, Itabashi-ku
  - Research Site, Kagoshima
  - Research Site, Kahoku-gun
  - Research Site, Kishiwada-shi
  - Research Site, Kobe
  - Research Site, Kyoto
  - Research Site, Maebashi
  - Research Site, Morioka
  - Research Site, Naka-gun
  - Research Site, Sagamihara-shi
  - Research Site, Sakaide-shi
  - Research Site, Sapporo
  - Research Site, Sumida-ku
  - Research Site, Takatsuki-shi
  - Research Site, Tomakomai-shi
  - Research Site, Wakayama
  - Research Site, Yokohama
- Mexico (7):
  - Research Site, Culiacán
  - Research Site, Guadalajara
  - Research Site, México
  - Research Site, Morelia
  - Research Site, Querétaro City
  - Research Site, Tampico
  - Research Site, Villahermosa
- Philippines (3):
  - Research Site, Iloilo City
  - Research Site, Lipa City
  - Research Site, Quezon City
- Poland (3):
  - Research Site, Lodz
  - Research Site, Wroclaw
  - Research Site, Zabrze
- Russia (5):
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Saint Petersburg
  - Research Site, Vladikavkaz
  - Research Site, Yekaterinburg
- South Korea (4):
  - Research Site, Bucheon-si
  - Research Site, Incheon
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (5):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Pamplona
  - Research Site, Sagunto(Valencia)
  - Research Site, Santander
- United Kingdom (2):
  - Research Site, Leicester
  - Research Site, Manchester

REFERENCES:
- [Background] Brightling CE, Chanez P, Leigh R, O'Byrne PM, Korn S, She D, May RD, Streicher K, Ranade K, Piper E. Efficacy and safety of tralokinumab in patients with severe uncontrolled asthma: a randomised, double-blind, placebo-controlled, phase 2b trial. Lancet Respir Med. 2015 Sep;3(9):692-701. doi: 10.1016/S2213-2600(15)00197-6. Epub 2015 Jul 28. PMID 26231288
- [Derived] Baverel PG, White N, Vicini P, Karlsson MO, Agoram B. Dose-Exposure-Response Relationship of the Investigational Anti-Interleukin-13 Monoclonal Antibody Tralokinumab in Patients With Severe, Uncontrolled Asthma. Clin Pharmacol Ther. 2018 May;103(5):826-835. doi: 10.1002/cpt.803. Epub 2017 Sep 28. PMID 28758192
- See also: CD-RI-CAT-354-1049 Redacted Protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=51&filename=CAT-354_CP1049_Protocol_Legal%20IP_Redacted_02Sep14.pdf
- See also: CD-RI-CAT-354-1049 SAP — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=51&filename=CAT-354_CP1049_SAP_08Aug14.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 689 participants were screened, out of which 452 participants were randomized into this study
Period: Overall Study
Arm/Group | Placebo, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2W - Cohort 1 | Placebo, Q2/4W - Cohort 2 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Started | 76 | 150 | 75 | 151
Completed | 67 | 135 | 67 | 129
Not Completed | 9 | 15 | 8 | 22
Not completed — Withdrawal by Subject | 7 | 10 | 7 | 13
Not completed — Death | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Other | 2 | 5 | 1 | 6

BASELINE CHARACTERISTICS:
Population: The intention-to-treat (ITT) population included all participants who were randomized into the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2W - Cohort 1 | Placebo, Q2/4W - Cohort 2 | Tralokinumab 300 mg, Q2/4W - Cohort 2 | Total
Number analyzed (Participants) | 76 | 150 | 75 | 151 | 452
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (12.1) | 49.7 (12.2) | 51.7 (13.6) | 50.5 (11.8) | 50.1 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 100 | 46 | 100 | 297
  Male | 25 | 50 | 29 | 51 | 155

OUTCOME MEASURES:

1. Primary Outcome: Annual Asthma Exacerbation Rate (AER)
Description: Annualized AER was assessed based on AER data up to Week 53. An asthma exacerbation defined as a progressive increase of asthma symptoms that does not resolve after the initiation of rescue medications and remains troublesome for the participant resulting in either 1) use of systemic corticosteroids or increase of a stable systemic maintenance dose for a duration of at least 3 consecutive days as prescribed or administered by the investigator or healthcare provider; or 2) participant initiation of systemic corticosteroids for a duration of at least 3 consecutive days. An asthma exacerbation event was considered resolved 7 days after the last dose of oral corticosteroids (OCS) is administered (10 days after administration of an injectable corticosteroid). Courses of corticosteroids initiated after this time period were considered a separate new asthma exacerbation. Data were summarized together for 'Placebo, Q2W' and 'Placebo, Q2/4W' arms.
Time Frame: Week 1 up to Week 53
Population: The intent-to-treat (ITT) population included all participants who were randomized into the study.
Measure: Number (95% Confidence Interval); unit: AER events/person-year
Groups:
- Placebo Total: Participants who received matching placebo subcutaneous injection every 2 weeks (Q2W) for a total of 26 doses up to 50 weeks, and participants who received matching placebo subcutaneous injection every 2 weeks (Q2W) for 12 weeks followed by every 4 weeks (Q4W) for 38 weeks (Q2/4W) for a total of 16 doses.
Arm/Group | Placebo Total | Tralokinumab 300 mg, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Number analyzed (Participants) | 151 | 150 | 151
AER events/person-year | 0.90 [0.75 to 1.08] | 0.91 [0.76 to 1.08] | 0.97 [0.81 to 1.14]
Statistical Analysis 1: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; The 95 percent (%) confidence interval (CI) for rate ratio were estimated from the Poisson regression with treatment group, age, gender, number of exacerbations in past year (2 versus [vs] more than [>] 2 but less than or equal to [=<] 6), atopic asthma status (atopic/non-atopic), chronic oral corticosteroid (OCS) use (presence vs absence) and geographical region as the covariates; Test type: Superiority or Other; p = 0.709, Poisson regression; Rate Ratio = 0.94, 95% CI 2-sided [0.67 to 1.31]
Statistical Analysis 2: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; The 95% CI for rate ratio were estimated from the Poisson regression with treatment group, age, gender, number of exacerbations in past year (2 vs > 2 but =< 6), atopic asthma status (atopic/non-atopic), chronic OCS use (presence vs absence) and geographical region as the covariates; Test type: Superiority or Other; p = 0.904, Poisson regression; Rate Ratio = 1.02, 95% CI 2-sided [0.71 to 1.46]

2. Secondary Outcome: Mean Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) at Week 53
Description: Pre- and post-bronchodilator FEV1 at clinic visits (morning) were measured. FEV1 was the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration. Data were summarized together for 'Placebo, Q2W' and 'Placebo, Q2/4W' arms.
Time Frame: Baseline and Week 53
Population: The ITT population included all participants who were randomized into the study. Here "n" signifies participants who were evaluable for this measure for the specified time point for each arm, respectively.
Measure: Mean (Standard Error); unit: liters
Arm/Group | Placebo Total | Tralokinumab 300 mg, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Number analyzed (Participants) | 151 | 150 | 151
liters
  Pre-bronchodilator: Baseline (n=147,146,146) | 1.926 (0.050) | 1.922 (0.056) | 1.934 (0.059)
  Post-bronchodilator: Baseline (n=147,141,146) | 2.153 (0.053) | 2.094 (0.061) | 2.110 (0.061)
  Pre-bronchodilator: Week 53 (n=125,130,122) | 0.018 (0.035) | 0.128 (0.032) | 0.032 (0.026)
  Post-bronchodilator: Week 53 (n=125,126,120) | -0.058 (0.027) | 0.085 (0.029) | -0.009 (0.025)

3. Secondary Outcome: Mean Change From Baseline in Forced Expiratory Volume in 6 Second (FEV6) at Week 53
Description: Pre- and post-bronchodilator FEV6 at clinic visits (morning) were measured. FEV6 was the maximal volume of air exhaled in the six second of a forced expiration from a position of full inspiration. Data were summarized together for 'Placebo, Q2W' and 'Placebo, Q2/4W' arms.
Time Frame: Baseline and Week 53
Population: as for outcome 2
Measure: Mean (Standard Error); unit: liters
Arm/Group | Placebo Total | Tralokinumab 300 mg, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Number analyzed (Participants) | 151 | 150 | 151
liters
  Pre-bronchodilator: Baseline (n=147,146,146) | 2.830 (0.064) | 2.809 (0.072) | 2.827 (0.074)
  Post-bronchodilator: Baseline (n=147,141,146) | 3.055 (0.067) | 2.981 (0.075) | 2.980 (0.076)
  Pre-bronchodilator: Week 53 (n=125,130,122) | 0.007 (0.036) | 0.117 (0.037) | 0.003 (0.031)
  Post-bronchodilator: Week 53 (n=125,126,120) | -0.057 (0.030) | 0.060 (0.033) | -0.024 (0.029)

4. Secondary Outcome: Mean Change From Baseline in Forced Vital Capacity (FVC) at Week 53
Description: Pre- and post-bronchodilator FVC at clinic visits (morning) were measured. FVC was the volume of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. Data were summarized together for 'Placebo, Q2W' and 'Placebo, Q2/4W' arms.
Time Frame: Baseline and Week 53
Population: as for outcome 2
Measure: Mean (Standard Error); unit: liters
Arm/Group | Placebo Total | Tralokinumab 300 mg, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Number analyzed (Participants) | 151 | 150 | 151
liters
  Pre-bronchodilator: Baseline (n=147,146,146) | 3.003 (0.069) | 2.955 (0.075) | 2.993 (0.079)
  Post-bronchodilator: Baseline (n=147,141,146) | 3.225 (0.072) | 3.133 (0.078) | 3.125 (0.080)
  Pre-bronchodilator: Week 53 (n=125,130,122) | -0.001 (0.039) | 0.110 (0.042) | -0.018 (0.032)
  Post-bronchodilator: Week 53 (n=125,126,120) | -0.071 (0.032) | 0.045 (0.034) | -0.030 (0.031)

5. Secondary Outcome: Mean Change From Baseline in Ratio of Forced Expiratory Volume in 1 Second (FEV1)/Forced Vital Capacity (FVC) at Week 53
Description: Pre- and post-bronchodilator FEV1 and FVC at clinic visits (morning) were measured. FEV1 was the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration. FVC was the volume of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. Ratio of FEV1/FVC was analysed. Data were summarized together for 'Placebo, Q2W' and 'Placebo, Q2/4W' arms.
Time Frame: Baseline and Week 53
Population: as for outcome 2
Measure: Mean (Standard Error); unit: percentage of ratio
Arm/Group | Placebo Total | Tralokinumab 300 mg, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Number analyzed (Participants) | 151 | 150 | 151
percentage of ratio
  Pre-bronchodilator: Baseline (n=147,146,146) | 64.508 (0.986) | 65.071 (1.013) | 65.008 (1.009)
  Post-bronchodilator: Baseline (n=147,141,146) | 67.152 (0.997) | 66.831 (1.056) | 67.883 (1.010)
  Pre-bronchodilator: Week 53 (n=125,130,122) | 0.320 (0.685) | 1.695 (0.517) | 1.155 (0.527)
  Post-bronchodilator: Week 53 (n=125,126,120) | -0.512 (0.513) | 1.593 (0.563) | 0.032 (0.484)

6. Secondary Outcome: Mean Change From Baseline in Inspiratory Capacity (IC) at Week 53
Description: Pre- and post-bronchodilator IC at clinic visits (morning) were measured. IC was measured by spirometry. Data were summarized together for 'Placebo, Q2W' and 'Placebo, Q2/4W' arms.
Time Frame: Baseline and Week 53
Population: as for outcome 2
Measure: Mean (Standard Error); unit: liters
Arm/Group | Placebo Total | Tralokinumab 300 mg, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Number analyzed (Participants) | 151 | 150 | 151
liters
  Pre-bronchodilator: Baseline (n=140,138,143) | 0.022 (0.001) | 0.023 (0.001) | 0.023 (0.001)
  Post-bronchodilator: Baseline (n=140,133,135) | 0.024 (0.001) | 0.024 (0.001) | 0.024 (0.001)
  Pre-bronchodilator: Week 53 (n=108,109,103) | 0.001 (0.001) | 0.000 (0.000) | 0.001 (0.001)
  Post-bronchodilator: Week 53 (n=108,109,104) | 0.000 (0.001) | 0.001 (0.001) | 0.000 (0.001)

7. Secondary Outcome: Mean Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) at Week 53 at Home
Description: Pre- and post-bronchodilator FEV1 at home (morning and evening) were measured. FEV1 was the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration. Data were summarized together for 'Placebo, Q2W' and 'Placebo, Q2/4W' arms.
Time Frame: Day 1 - Day 7 (Baseline) and Day 365 - Day 371 (Week 53)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: liters
Arm/Group | Placebo Total | Tralokinumab 300 mg, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Number analyzed (Participants) | 151 | 150 | 151
liters
  Day 1-7: Morning (n=151,149,149) | 1.63 (0.05) | 1.61 (0.05) | 1.66 (0.05)
  Change at Day 365-371: Morning (n=124,119,114) | -0.12 (0.06) | 0.01 (0.04) | -0.07 (0.06)
  Day 1-7: Evening (n=149,147,148) | 1.61 (0.05) | 1.68 (0.05) | 1.65 (0.05)
  Change at Day 365-371: Evening (n=120,116,112) | -0.08 (0.05) | -0.08 (0.05) | -0.12 (0.05)

8. Secondary Outcome: Mean Change From Baseline in Peak Expiratory Flow (PEF) at Week 53 at Home
Description: The PEF is a participant's maximum speed of expiration, as measured with a peak flow meter. Peak flow testing for PEF was performed at home (morning and evening) while sitting or standing prior to using any medication (if needed) for asthma. Data were summarized together for 'Placebo, Q2W' and 'Placebo, Q2/4W' arms.
Time Frame: Day 1 - Day 7 (Baseline) and Day 365 - Day 371 (Week 53)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: liters per minute
Arm/Group | Placebo Total | Tralokinumab 300 mg, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Number analyzed (Participants) | 151 | 150 | 151
liters per minute
  Day 1-7: Morning (n=151,149,149) | 273.7 (8.7) | 271.0 (9.7) | 281.2 (9.9)
  Change at Day 365-371: Morning (n=124,119,114) | -23.1 (8.8) | -8.0 (7.9) | -24.0 (9.6)
  Day 1-7: Evening (n=149,147,148) | 276.0 (8.9) | 287.6 (9.9) | 283.8 (10.0)
  Change at Day 365-371: Evening (n=120,116,112) | -16.4 (8.7) | -27.0 (8.2) | -36.5 (8.8)

9. Secondary Outcome: Change From Baseline in Mean Asthma Control Questionnaire (6-items) (ACQ-6) Score at Week 53
Description: Asthma Control Questionnaire (ACQ) is a participant-reported questionnaire to assess the asthma control with 6 items assessing night-time waking, symptoms on waking, activity limitation, shortness of breath, wheeze, and rescue short-acting beta agonist use. Each item was rated on a 7-point Likert scale ranging from 0 (no impairment) to 6 (maximum impairment). Overall ACQ score was the mean of the 6 item scores with a score range of 0 (well controlled) to 6 (extremely poor controlled). Data collected on Day 1 prior to dosing was considered as baseline. Results were reported for overall ACQ score. Data were summarized together for 'Placebo, Q2W' and 'Placebo, Q2/4W' arms.
Time Frame: Baseline and Week 53
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Total | Tralokinumab 300 mg, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Number analyzed (Participants) | 151 | 150 | 151
units on a scale
  Baseline (n=149,147,148) | 2.52 (0.07) | 2.59 (0.09) | 2.54 (0.08)
  Change at Week 53 (n=118,115,112) | -0.82 (0.10) | -1.02 (0.10) | -0.93 (0.11)

10. Secondary Outcome: Change From Baseline in Asthma Quality of Life Questionnaire Standardized Version (AQLQ[S]) Score at Week 53
Description: AQLQ: a 32-item questionnaire evaluating quality of life of participants with asthma including 4 domains (symptoms, activity limitations, emotional function, and environmental stimuli). Participants were asked to recall their experiences during the previous 2 weeks and to score each of the 32 questions on a 7-point scale ranging from 7 (no impairment) to 1 (severe impairment). The overall score was calculated as the mean response to all questions. The 4 domain scores were the means of the responses to the questions in each of the domains. Overall AQLQ score and 4 domain scores ranged from 7 (no impairment) to 1 (severe impairment). Data were summarized together for 'Placebo, Q2W' and 'Placebo, Q2/4W' arms.
Time Frame: Baseline and Week 53
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Total | Tralokinumab 300 mg, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Number analyzed (Participants) | 151 | 150 | 151
units on a scale
  Baseline: Overall (n=147,142,141) | 4.05 (0.09) | 3.98 (0.09) | 4.08 (0.09)
  Week 53: Overall (n=107,109,101) | 0.85 (0.10) | 1.04 (0.10) | 1.00 (0.12)
  Baseline: Symptoms (n=147,142,141) | 4.10 (0.09) | 4.03 (0.09) | 4.13 (0.09)
  Week 53: Symptoms (n=107,109,101) | 0.85 (0.11) | 1.14 (0.12) | 1.05 (0.13)
  Baseline: Activity limitation (n=147,142,141) | 4.04 (0.08) | 4.04 (0.09) | 4.13 (0.09)
  Week 53: Activity limitation (n=107,109,101) | 0.81 (0.10) | 0.96 (0.10) | 0.93 (0.12)
  Baseline: Emotional Function (n=147,142,141) | 4.14 (0.12) | 3.91 (0.12) | 4.02 (0.11)
  Week 53: Emotional Function (n=107,109,101) | 0.89 (0.12) | 1.10 (0.12) | 1.09 (0.15)
  Baseline: Environmental stimuli (n=147,142,141) | 3.80 (0.11) | 3.76 (0.12) | 3.89 (0.12)
  Week 53: Environmental stimuli (n=107,109,101) | 0.88 (0.13) | 0.86 (0.14) | 0.97 (0.14)

11. Secondary Outcome: Number of Participants With European Quality of Life 5 Dimensions (EQ-5D) Scores at Week 53
Description: The utility-based EQ-5D questionnaire comprises of two parts and provides a generic measure of health for clinical and economic appraisal. The health state valuation was the summary score of mobility, self-care, usual activities, pain/discomfort and anxiety/depression on a 3 category scale (no problem, moderate problem, severe problems) that reflects increasing levels of difficulty. The minimum possible value is 5 (one point for each dimension) and the maximum possible values is 15 (3 points for each dimension). Data were summarized together for 'Placebo, Q2W' and 'Placebo, Q2/4W' arms.
Time Frame: Week 53
Population: The ITT population included all participants who were randomized into the study.
Measure: Number; unit: participants
Arm/Group | Placebo Total | Tralokinumab 300 mg, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Number analyzed (Participants) | 151 | 150 | 151
participants
  Mobility - No problem | 107 (0.10) | 118 (0.10) | 106 (0.12)
  Mobility - Moderate problem | 26 (0.12) | 18 (0.12) | 23 (0.11)
  Mobility - Severe Problem | 1 (0.12) | 0 (0.12) | 1 (0.15)
  Mobility - Missing | 17 (0.13) | 14 (0.14) | 21 (0.14)
  Self-care - No Problem | 122 | 127 | 122
  Self-care - Moderate Problem | 12 | 9 | 7
  Self-care - Severe Problem | 0 | 0 | 1
  Self-care - Missing | 17 | 14 | 21
  Usual activities - No Problem | 89 | 106 | 100
  Usual activities - Moderate Problem | 43 | 30 | 30
  Usual activities - Severe Problem | 2 | 0 | 0
  Usual activities - Missing | 17 | 14 | 21
  Pain/discomfort - No problem | 84 | 100 | 77
  Pain/discomfort - Moderate problem | 46 | 34 | 51
  Pain/discomfort - Severe problem | 4 | 2 | 2
  Pain/discomfort - Missing | 17 | 14 | 21
  Anxiety/depression - No problem | 102 | 101 | 101
  Anxiety/depression - Moderate problem | 29 | 34 | 29
  Anxiety/depression - Severe problem | 3 | 1 | 0
  Anxiety/depression - Missing | 17 | 14 | 21

12. Secondary Outcome: Change From Baseline in European Quality of Life 5 Dimensions (EQ-5D) Visual Analog Scale (VAS) at Week 53
Description: The utility-based EQ-5D questionnaire comprises of two parts and provides a generic measure of health for clinical and economic appraisal. The EQ-5D VAS was measured from 0 (worst imaginable health state) to 100 (best imaginable health state). Data were summarized together for 'Placebo, Q2W' and 'Placebo, Q2/4W' arms.
Time Frame: Baseline and Week 53
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Total | Tralokinumab 300 mg, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Number analyzed (Participants) | 130 | 136 | 127
units on a scale | 8.4 (1.6) | 9.3 (1.9) | 7.3 (1.8)

13. Secondary Outcome: Change From Baseline in Assessing Symptoms of Moderate-to-severe Asthma (ASMA) at Week 53
Description: There were 3 symptom questions in the ASMA diary: daytime frequency (question 1), daytime severity (question 2) and nighttime severity (question 6). All symptom questions were scored from 0 to 4 averaged, where a higher score indicated greater frequency or severity. Daily Asthma symptom scores were averaged weekly for participants with at least 4 non-missing records each week. The baseline score was calculated from Day -7 to Day -1. Data were summarized together for 'Placebo, Q2W' and 'Placebo, Q2/4W' arms.
Time Frame: Day -7 - Day -1 (Baseline) and Day 365 - Day 371 (Week 53)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Total | Tralokinumab 300 mg, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Number analyzed (Participants) | 151 | 150 | 151
units on a scale
  Day -7 - Day -1 (Baseline) (n=151,147,145) | 1.60 (0.71) | 1.49 (0.77) | 1.56 (0.69)
  Change at Day 365 - Day 371 (n=113,108,108) | -0.43 (0.75) | -0.42 (0.73) | -0.49 (0.78)

14. Secondary Outcome: Change From Baseline in Rescue Medication Use at Week 53
Description: Rescue medication use was collected from 3 questions: daytime use in response to symptoms (question 3), daytime prophylactic use (question 4) and nighttime use (question 7). Rescue medication use questions were first assessed using a dichotomous response option (YES/NO). If the participants reported YES, there was a subsequent question about the number of times rescue medication was used (questions 3a, 4a, and 7a). Daily average scores were summarized each week for all participants with at least 4 non-missing records each week. Days with no reported rescue medication use were represented as 0 and included in the calculation with participants who reported yes and completed questions 3a, 4a and 7a. The baseline scores were calculated from Day -7 to Day -1. Data were summarized together for 'Placebo, Q2W' and 'Placebo, Q2/4W' arms.
Time Frame: Day -7 - Day -1 (Baseline) and Day 365 - Day 371 (Week 53)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: use per day
Arm/Group | Placebo Total | Tralokinumab 300 mg, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Number analyzed (Participants) | 151 | 150 | 151
use per day
  Day -7 - Day -1 (Baseline) (n=151,147,145) | 2.56 (2.73) | 2.77 (3.78) | 2.38 (2.58)
  Change at Day 365 - Day 371 (n=113,108,108) | -0.86 (2.20) | -0.77 (2.59) | -1.02 (2.30)

15. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between administration of study drug and up to Week 75 that were absent before treatment or that worsened relative to pre-treatment state. Data were summarized together for 'Placebo, Q2W' and 'Placebo, Q2/4W' arms.
Time Frame: Baseline and Week 75
Population: The safety population included all participants who received any investigational product and had safety data available for analysis.
Measure: Number; unit: participants
Arm/Group | Placebo Total | Tralokinumab 300 mg, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Number analyzed (Participants) | 151 | 150 | 151
participants
  TEAEs | 129 (17.12) | 134 (19.83) | 128 (16.98)
  TESAEs | 21 (1.6) | 18 (1.9) | 25 (1.8)

16. Secondary Outcome: Observed Serum Tralokinumab Concentration at Week 53
Description: Tralokinumab concentrations that were below limit of quantification (LOQ) of the pharmacokinetic (PK) assay (LOQ = 0.500 microgram per milliliter [mcg/mL]) were replaced by LOQ/2 = 0.250 mcg/mL; results were reported to 3 significant figures level of precision. Observed serum tralokinumab concentration at Week 53 was reported.
Time Frame: Week 53
Population: The PK population included all participants who received at least one dose of tralokinumab and had at least one quantifiable PK observation. Here "N" signifies participants who were evaluable for this measure for the specified time point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: microgram per milliliter
Arm/Group | Tralokinumab 300 mg, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Number analyzed (Participants) | 136 | 128
microgram per milliliter | 71.3 (34.2) | 25.8 (11.8)

17. Secondary Outcome: Percentage of Participants With Anti-Drug Antibodies (ADA) to Tralokinumab
Description: Immunogenicity assessment included determination of anti-drug (tralokinumab) antibodies in serum samples. ADA positive was defined as a titer greater than or equal to (>=13) at any point in the study. Data were summarized together for 'Placebo, Q2W' and 'Placebo, Q2/4W' arms.
Time Frame: Baseline and Week 75
Population: as for outcome 16
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Total | Tralokinumab 300 mg, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Number analyzed (Participants) | 151 | 150 | 151
percentage of participants
  Baseline (Week 1) (n=151,150,151) | 1.3 (17.12) | 0.67 (19.83) | 1.3 (16.98)
  Week 75 (n=151,150,150) | 3.3 | 0.0 | 4.0

18. Secondary Outcome: Severe Annual Asthma Exacerbation Rate (AER)
Description: Severe annualized AER was assessed based on AER data up to Week 53. Annualized AER was assessed based on AER data up to Week 53. An asthma exacerbation defined as a progressive increase of asthma symptoms that does not resolve after the initiation of rescue medications and remains troublesome for the participant resulting in either 1) use of systemic corticosteroids or increase of a stable systemic maintenance dose for a duration of at least 3 consecutive days as prescribed or administered by the investigator; or 2) participant initiation of systemic corticosteroids for a duration of at least 3 consecutive days. An asthma exacerbation event was considered resolved 7 days after the last dose of oral corticosteroids is administered (10 days after an injectable corticosteroid). Courses of corticosteroids initiated after this time period were considered a separate new asthma exacerbation. Data were summarized together for 'Placebo, Q2W' and 'Placebo, Q2/4W' arms.
Time Frame: Week 1 up to Week 53
Population: The ITT population included all participants who were randomized into the study.
Measure: Number (95% Confidence Interval); unit: AER events/person-year
Arm/Group | Placebo Total | Tralokinumab 300 mg, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Number analyzed (Participants) | 151 | 150 | 151
AER events/person-year | 0.17 [0.10 to 0.25] | 0.11 [0.06 to 0.17] | 0.10 [0.05 to 0.17]
Statistical Analysis 1: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; The 95% CI for rate ratio were estimated from the Poisson regression with treatment group, age, gender, number of exacerbations in past year (2 vs >2 but =<6), atopic asthma status (atopic/non-atopic), chronic OCS use (presence vs absence) and geographical region as the covariates; Test type: Superiority or Other; p = 0.293, Poisson regression; Rate Ratio = 0.62, 95% CI 2-sided [0.26 to 1.51]
Statistical Analysis 2: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; [analysis description as in outcome 18, analysis 1]; Test type: Superiority or Other; p = 0.270, Poisson regression; Rate Ratio = 0.62, 95% CI 2-sided [0.27 to 1.44]

19. Secondary Outcome: Time to First Exacerbation Through Week 53
Description: Data were summarized together for 'Placebo, Q2W' and 'Placebo, Q2/4W' arms.
Time Frame: Week 1 up to Week 53
Population: The ITT population included all participants who were randomized into the study.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo Total | Tralokinumab 300 mg, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Number analyzed (Participants) | 151 | 150 | 151
days | NA [NA to NA] — The median and lower and upper limits of the 95% Confidence Interval were incalculable due to an insufficient number of events. | NA [NA to NA] — The median and lower and upper limits of the 95% Confidence Interval were incalculable due to an insufficient number of events. | NA [NA to NA] — The median and lower and upper limits of the 95% Confidence Interval were incalculable due to an insufficient number of events.
Statistical Analysis 1: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Test type: Superiority or Other; p = 0.257, Regression, Cox; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.57 to 1.16]
Statistical Analysis 2: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Test type: Superiority or Other; p = 0.225, Regression, Cox; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.56 to 1.15]

20. Secondary Outcome: Time to First Severe Exacerbation Through Week 53
Description: Data were summarized together for 'Placebo, Q2W' and 'Placebo, Q2/4W' arms.
Time Frame: Week 1 up to Week 53
Population: The ITT population included all participants who were randomized into the study.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo Total | Tralokinumab 300 mg, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Number analyzed (Participants) | 151 | 150 | 151
days | NA [NA to NA] — The median and lower and upper limits of the 95% Confidence Interval were incalculable due to an insufficient number of events. | NA [NA to NA] — The median and lower and upper limits of the 95% Confidence Interval were incalculable due to an insufficient number of events. | NA [NA to NA] — The median and lower and upper limits of the 95% Confidence Interval were incalculable due to an insufficient number of events.
Statistical Analysis 1: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Test type: Superiority or Other; p = 0.538, Regression, Cox; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.37 to 1.68]
Statistical Analysis 2: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Test type: Superiority or Other; p = 0.561, Regression, Cox; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.37 to 1.71]

21. Secondary Outcome: Annual Asthma Exacerbation Rate (AER) by Baseline Serum Periostin
Description: Annualized AER was assessed based on AER data up to Week 53. An asthma exacerbation defined as a progressive increase of asthma symptoms that does not resolve after the initiation of rescue medications and remains troublesome for the participant resulting in either 1) use of systemic corticosteroids or increase of a stable systemic maintenance dose for a duration of at least 3 consecutive days as prescribed; or 2) participant initiation of systemic corticosteroids for a duration of at least 3 consecutive days. It was considered resolved 7 days after the last dose of OCS administered (10 days after an injectable corticosteroid). Courses of corticosteroids initiated after this time period were considered a separate new asthma exacerbation. AER was evaluated by subgroup baseline serum periostin greater than or equal to (>=) or less than (<) median, >= or < 25th percentile and >= or < 75th percentile. Data were summarized together for 'Placebo, Q2W' and 'Placebo, Q2/4W' arms.
Time Frame: Week 1 up to Week 53
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: AER events/person-year
Arm/Group | Placebo Total | Tralokinumab 300 mg, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Number analyzed (Participants) | 151 | 150 | 151
AER events/person-year
  >= median (n=67,81,79) | 1.13 [0.88 to 1.43] | 0.85 [0.65 to 1.08] | 1.27 [1.03 to 1.55]
  < median (n=84,69,71) | 0.73 [0.55 to 0.95] | 0.98 [0.76 to 1.25] | 0.63 [0.45 to 0.85]
  >= 25th Percentile (n=105,115,119) | 0.94 [0.75 to 1.15] | 0.84 [0.67 to 1.03] | 1.05 [0.87 to 1.25]
  < 25th Percentile (n=46,35,31) | 0.83 [0.58 to 1.16] | 1.14 [0.81 to 1.56] | 0.65 [0.38 to 1.05]
  >= 75th Percentile (n=32,43,39) | 1.13 [0.76 to 1.60] | 0.91 [0.65 to 1.25] | 2.03 [1.60 to 2.55]
  < 75th Percentile (n=119,107,111) | 0.85 [0.69 to 1.04] | 0.91 [0.73 to 1.11] | 0.60 [0.46 to 0.77]
Statistical Analysis 1: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline serum periostin >= median; Test type: Superiority or Other; p = 0.190, Poisson regression; Rate Ratio = 0.73, 95% CI 2-sided [0.46 to 1.17] — The 95% CI for rate ratio were estimated from the Poisson regression with treatment group, age, gender, number of exacerbations in past year (2 vs >2 but =<6), atopic asthma status, chronic OCS use and geographical region as the covariates
Statistical Analysis 2: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline serum periostin >= median; Test type: Superiority or Other; p = 0.856, Poisson regression; Rate Ratio = 0.95, 95% CI 2-sided [0.56 to 1.61] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 3: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline serum periostin < median; Test type: Superiority or Other; p = 0.602, Poisson regression; Rate Ratio = 1.13, 95% CI 2-sided [0.71 to 1.81] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 4: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline serum periostin < median; Test type: Superiority or Other; p = 0.703, Poisson regression; Rate Ratio = 0.91, 95% CI 2-sided [0.55 to 1.50] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 5: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline serum periostin >= 25th Percentile; Test type: Superiority or Other; p = 0.455, Poisson regression; Rate Ratio = 0.86, 95% CI 2-sided [0.58 to 1.28] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 6: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline serum periostin >= 25th Percentile; Test type: Superiority or Other; p = 0.929, Poisson regression; Rate Ratio = 1.02, 95% CI 2-sided [0.66 to 1.57] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 7: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline serum periostin < 25th Percentile; Test type: Superiority or Other; p = 0.507, Poisson regression; Rate Ratio = 1.26, 95% CI 2-sided [0.63 to 2.51] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 8: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline serum periostin < 25th Percentile; Test type: Superiority or Other; p = 0.805, Poisson regression; Rate Ratio = 0.91, 95% CI 2-sided [0.44 to 1.89] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 9: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline serum periostin >= 75th Percentile; Test type: Superiority or Other; p = 0.716, Poisson regression; Rate Ratio = 0.88, 95% CI 2-sided [0.44 to 1.75] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 10: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline serum periostin >= 75th Percentile; Test type: Superiority or Other; p = 0.328, Poisson regression; Rate Ratio = 1.51, 95% CI 2-sided [0.66 to 3.43] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 11: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline serum periostin < 75th Percentile; Test type: Superiority or Other; p = 0.804, Poission regression; Rate Ratio = 0.95, 95% CI 2-sided [0.64 to 1.41] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 12: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline serum periostin < 75th Percentile; Test type: Superiority or Other; p = 0.088, Poisson regression; Rate Ratio = 0.70, 95% CI 2-sided [0.47 to 1.05] — [estimate comment as in outcome 21, analysis 1]

22. Secondary Outcome: Annual Asthma Exacerbation Rate (AER) by T-helper-2 (Th2) Status
Description: Annualized AER was assessed based on AER data up to Week 53. An asthma exacerbation defined as a progressive increase of asthma symptoms that does not resolve after the initiation of rescue medications and remains troublesome for the participant resulting in either 1) use of systemic corticosteroids or increase of a stable systemic maintenance dose for a duration of at least 3 consecutive days as prescribed; or 2) participant initiation of systemic corticosteroids for a duration of at least 3 consecutive days. AER was evaluated by subgroup Th2 status. Th2-high included those participants who had immunoglobulin E (IgE) >100 international unit per milliliter (IU/mL) and blood eosinophils >= 0.14 * 10 power 9 per Liter. Th2 low would include those participants who do not meet Th2 high status. Data were summarized together for 'Placebo, Q2W' and 'Placebo, Q2/4W' arms.
Time Frame: Week 1 up to Week 53
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: AER events/person-year
Arm/Group | Placebo Total | Tralokinumab 300 mg, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Number analyzed (Participants) | 151 | 150 | 151
AER events/person-year
  Th2 high (n=70,74,67) | 0.96 [0.74 to 1.23] | 0.94 [0.73 to 1.20] | 1.09 [0.85 to 1.39]
  Th2 Low (n=73,61,72) | 0.90 [0.69 to 1.16] | 0.88 [0.66 to 1.16] | 0.85 [0.64 to 1.11]
Statistical Analysis 1: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Th2 high; Test type: Superiority or Other; p = 0.365, Poisson regression; Rate Ratio = 0.80, 95% CI 2-sided [0.50 to 1.29] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 2: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Th2 high; Test type: Superiority or Other; p = 0.922, Poisson regression; Rate Ratio = 0.97, 95% CI 2-sided [0.56 to 1.68] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 3: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Th2 Low; Test type: Superiority or Other; p = 0.685, Poisson regression; Rate Ratio = 1.11, 95% CI 2-sided [0.67 to 1.84] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 4: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Th2 Low; Test type: Superiority or Other; p = 0.813, Poisson regression; Rate Ratio = 1.06, 95% CI 2-sided [0.66 to 1.70] — [estimate comment as in outcome 21, analysis 1]

23. Secondary Outcome: Annual Asthma Exacerbation Rate (AER) by Baseline Peripheral Blood Eosinophil Count
Description: Annualized AER was assessed based on AER data up to Week 53. An asthma exacerbation defined as a progressive increase of asthma symptoms that does not resolve after the initiation of rescue medications and remains troublesome for the participant resulting in either 1) use of systemic corticosteroids or increase of a stable systemic maintenance dose for a duration of at least 3 consecutive days as prescribed; or 2) participant initiation of systemic corticosteroids for a duration of at least 3 consecutive days. It was considered resolved 7 days after the last dose of OCS administered (10 days after an injectable corticosteroid). Courses of corticosteroids initiated after this time period were considered a separate new asthma exacerbation. AER evaluated by subgroups baseline peripheral blood eosinophil counts. Data were summarized together for 'Placebo, Q2W' and 'Placebo, Q2/4W' arms.
Time Frame: Week 1 up to Week 53
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: AER events/person-year
Arm/Group | Placebo Total | Tralokinumab 300 mg, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Number analyzed (Participants) | 151 | 150 | 151
AER events/person-year
  >= 150 cells/mcgL (n=95,104,92) | 0.95 [0.76 to 1.18] | 0.84 [0.66 to 1.04] | 0.96 [0.77 to 1.19]
  < 150 cells/mcgL (n=48,38,52) | 0.90 [0.64 to 1.22] | 1.09 [0.78 to 1.48] | 0.95 [0.69 to 1.27]
  >= 300 cells/mcgL (n=54,60,50) | 1.00 [0.74 to 1.32] | 1.01 [0.76 to 1.31] | 1.56 [1.23 to 1.97]
  < 300 cells/mcgL (n=89,82,94) | 0.89 [0.70 to 1.12] | 0.83 [0.64 to 1.06] | 0.63 [0.47 to 0.82]
Statistical Analysis 1: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline eosinophil count >=150 cells/mcgL; Test type: Superiority or Other; p = 0.335, Poisson regression; Rate Ratio = 0.82, 95% CI 2-sided [0.56 to 1.22] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 2: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline eosinophil count >=150 cells/mcgL; Test type: Superiority or Other; p = 0.586, Poisson regression; Rate Ratio = 0.88, 95% CI 2-sided [0.54 to 1.41] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 3: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline eosinophil count <150 cells/mcgL; Test type: Superiority or Other; p = 0.331, Poisson regression; Rate Ratio = 1.36, 95% CI 2-sided [0.73 to 2.52] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 4: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline eosinophil count <150 cells/mcgL; Test type: Superiority or Other; p = 0.311, Poisson regression; Rate Ratio = 1.41, 95% CI 2-sided [0.73 to 2.71] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 5: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline eosinophil count >=300 cells/mcgL; Test type: Superiority or Other; p = 0.414, Poisson regression; Rate Ratio = 0.81, 95% CI 2-sided [0.48 to 1.35] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 6: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline eosinophil count >=300 cells/mcgL; Test type: Superiority or Other; p = 0.463, Poisson regression; Rate Ratio = 1.26, 95% CI 2-sided [0.68 to 2.36] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 7: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline eosinophil count <300 cells/mcgL; Test type: Superiority or Other; p = 0.793, Poisson regression; Rate Ratio = 1.06, 95% CI 2-sided [0.67 to 1.68] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 8: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline eosinophil count <300 cells/mcgL; Test type: Superiority or Other; p = 0.264, Poisson regression; Rate Ratio = 0.77, 95% CI 2-sided [0.49 to 1.22] — [estimate comment as in outcome 21, analysis 1]

24. Secondary Outcome: Annual Asthma Exacerbation Rate (AER) by Baseline FEV1 Reversibility
Description: Annualized AER was assessed based on AER data up to Week 53. An asthma exacerbation defined as a progressive increase of asthma symptoms that does not resolve after the initiation of rescue medications and remains troublesome for the participant resulting in either 1) use of systemic corticosteroids or increase of a stable systemic maintenance dose for a duration of at least 3 consecutive days as prescribed; or 2) participant initiation of systemic corticosteroids for a duration of at least 3 consecutive days. It was considered resolved 7 days after the last dose of OCS administered (10 days after an injectable corticosteroid). Courses of corticosteroids initiated after this time period were considered a separate new asthma exacerbation. AER evaluated by subgroup baseline FEV1 reversibility >=12% and <12%. Data were summarized together for 'Placebo, Q2W' and 'Placebo, Q2/4W' arms.
Time Frame: Week 1 up to Week 53
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: AER events/person-year
Arm/Group | Placebo Total | Tralokinumab 300 mg, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Number analyzed (Participants) | 151 | 150 | 151
AER events/person-year
  Reversibility >=12% (n=57,43,49) | 0.88 [0.65 to 1.18] | 0.68 [0.45 to 0.99] | 1.08 [0.80 to 1.42]
  Reversibility <12% (n=91,101,97) | 0.93 [0.73 to 1.16] | 0.99 [0.80 to 1.21] | 0.90 [0.71 to 1.12]
Statistical Analysis 1: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline FEV1 reversibility >=12%; Test type: Superiority or Other; p = 0.245, Poisson regression; Rate Ratio = 0.66, 95% CI 2-sided [0.33 to 1.32] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 2: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline FEV1 reversibility >=12%; Test type: Superiority or Other; p = 0.438, Poisson regression; Rate Ratio = 0.76, 95% CI 2-sided [0.37 to 1.54] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 3: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline FEV1 reversibility <12%; Test type: Superiority or Other; p = 0.947, Poisson regression; Rate Ratio = 1.01, 95% CI 2-sided [0.66 to 1.57] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 4: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline FEV1 reversibility <12%; Test type: Superiority or Other; p = 0.916, Poisson regression; Rate Ratio = 0.97, 95% CI 2-sided [0.59 to 1.59] — [estimate comment as in outcome 21, analysis 1]

25. Secondary Outcome: Annual Asthma Exacerbation Rate (AER) by Baseline FEV1% Predicted
Description: Annualized AER was assessed based on AER data up to Week 53. An asthma exacerbation defined as a progressive increase of asthma symptoms that does not resolve after the initiation of rescue medications and remains troublesome for the participant resulting in either 1) use of systemic corticosteroids or increase of a stable systemic maintenance dose for a duration of at least 3 consecutive days as prescribed; or 2) participant initiation of systemic corticosteroids for a duration of at least 3 consecutive days. It was considered resolved 7 days after the last dose of OCS administered (10 days after an injectable corticosteroid). Courses of corticosteroids initiated after this time period were considered a separate new asthma exacerbation. AER was evaluated by subgroup baseline FEV1% predicaed. Data were summarized together for 'Placebo, Q2W' and 'Placebo, Q2/4W' arms.
Time Frame: Week 1 up to Week 53
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: AER events/person-year
Arm/Group | Placebo Total | Tralokinumab 300 mg, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Number analyzed (Participants) | 151 | 150 | 151
AER events/person-year
  FEV1% Predicted <=60% (n=49,45,56) | 1.05 [0.77 to 1.40] | 0.95 [0.68 to 1.29] | 1.67 [1.34 to 2.07]
  FEV1% Predicted <=80% (n=119,109,105) | 0.93 [0.76 to 1.13] | 0.88 [0.71 to 1.08] | 1.13 [0.93 to 1.36]
Statistical Analysis 1: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline FEV1% predicted <=60%; Test type: Superiority or Other; p = 0.723, Poisson regression; Rate Ratio = 0.91, 95% CI 2-sided [0.52 to 1.56] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 2: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline FEV1% predicted <=60%; Test type: Superiority or Other; p = 0.852, Poisson regression; Rate Ratio = 1.06, 95% CI 2-sided [0.60 to 1.86] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 3: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline FEV1% predicted <=80%; Test type: Superiority or Other; p = 0.409, Poisson regression; Rate Ratio = 0.86, 95% CI 2-sided [0.60 to 1.23] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 4: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline FEV1% predicted <=80%; Test type: Superiority or Other; p = 0.744, Poisson regression; Rate Ratio = 1.07, 95% CI 2-sided [0.72 to 1.58] — [estimate comment as in outcome 21, analysis 1]

26. Secondary Outcome: Annual Asthma Exacerbation Rate (AER) by Asthma Exacerbations in the Past Year
Description: Annualized AER was assessed based on AER data up to Week 53. An asthma exacerbation defined as a progressive increase of asthma symptoms that does not resolve after the initiation of rescue medications and remains troublesome for the participant resulting in either 1) use of systemic corticosteroids or increase of a stable systemic maintenance dose for a duration of at least 3 consecutive days as prescribed; or 2) participant initiation of systemic corticosteroids for a duration of at least 3 consecutive days. It was considered resolved 7 days after the last dose of OCS administered (10 days after an injectable corticosteroid). Courses of corticosteroids initiated after this time period were considered a separate new asthma exacerbation. AER evaluated by subgroup as asthma exacerbations in the past year. Data were summarized together for 'Placebo, Q2W' and 'Placebo, Q2/4W' arms.
Time Frame: Week 1 up to Week 53
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: AER events/person-year
Arm/Group | Placebo Total | Tralokinumab 300 mg, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Number analyzed (Participants) | 151 | 150 | 151
AER events/person-year
  2 asthma exacerbations (n=97,96,95) | 0.62 [0.47 to 0.81] | 0.61 [0.45 to 0.79] | 0.45 [0.32 to 0.61]
  > 2 but < 6 asthma exacerbations (n=54,54,56) | 1.44 [1.12 to 1.82] | 1.42 [1.12 to 1.78] | 1.88 [1.52 to 2.30]
Statistical Analysis 1: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; 2 asthma exacerbations in the past year; Test type: Superiority or Other; p = 0.802, Poisson regression; Rate Ratio = 0.94, 95% CI 2-sided [0.58 to 1.52] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 2: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; 2 asthma exacerbations in the past year; Test type: Superiority or Other; p = 0.050, Poisson regression; Rate Ratio = 0.60, 95% CI 2-sided [0.36 to 1.00] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 3: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; > 2 but < 6 asthma exacerbations in the past year; Test type: Superiority or Other; p = 0.792, Poisson regression; Rate Ratio = 0.93, 95% CI 2-sided [0.56 to 1.56] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 4: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; > 2 but < 6 asthma exacerbations in the past year; Test type: Superiority or Other; p = 0.231, Poisson regression; Rate Ratio = 1.39, 95% CI 2-sided [0.81 to 2.38] — [estimate comment as in outcome 21, analysis 1]

27. Secondary Outcome: Severe Asthma Exacerbation Rate (AER) by Baseline Serum Periostin
Description: Severe AER was assessed based on AER data up to Week 53. Annualized AER was assessed based on AER data up to Week 53. An asthma exacerbation defined as a progressive increase of asthma symptoms that does not resolve after the initiation of rescue medications and remains troublesome for the participant resulting in either 1) use of systemic corticosteroids or increase of a stable systemic maintenance dose for a duration of at least 3 consecutive days as prescribed; or 2) participant initiation of systemic corticosteroids for a duration of at least 3 consecutive days. It was considered resolved 7 days after the last dose of OCS administered (10 days after an injectable corticosteroid). Courses of corticosteroids initiated after this time period were considered a separate new asthma exacerbation. Severe AER evaluated by subgroup baseline serum periostin. Data were summarized together for 'Placebo, Q2W' and 'Placebo, Q2/4W' arms.
Time Frame: Week 1 up to Week 53
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: AER events/person-year
Arm/Group | Placebo Total | Tralokinumab 300 mg, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Number analyzed (Participants) | 151 | 150 | 151
AER events/person-year
  >= median (n=67,81,79) | 0.25 [0.14 to 0.40] | 0.08 [0.03 to 0.17] | 0.12 [0.06 to 0.23]
  < median (n=84,69,71) | 0.10 [0.04 to 0.20] | 0.14 [0.06 to 0.26] | 0.08 [0.03 to 0.18]
Statistical Analysis 1: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline Serum Periostin >=Median; Test type: Superiority or Other; p = 0.046, Poisson regression; Rate Ratio = 0.25, 95% CI 2-sided [0.06 to 0.98] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 2: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline Serum Periostin >=Median; Test type: Superiority or Other; p = 0.197, Poisson regression; Rate Ratio = 0.47, 95% CI 2-sided [0.15 to 1.48] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 3: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline Serum Periostin < Median; Test type: Superiority or Other; p = 0.708, Poisson regression; Rate Ratio = 1.18, 95% CI 2-sided [0.50 to 2.79] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 4: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline Serum Periostin < Median; Test type: Superiority or Other; p = 0.594, Poisson regression; Rate Ratio = 1.31, 95% CI 2-sided [0.48 to 3.57] — [estimate comment as in outcome 21, analysis 1]

28. Secondary Outcome: Severe Asthma Exacerbation Rate (AER) by Baseline FEV1 Reversibility
Description: Severe AER was assessed based on AER data up to Week 53. Annualized AER was assessed based on AER data up to Week 53. An asthma exacerbation defined as a progressive increase of asthma symptoms that does not resolve after the initiation of rescue medications and remains troublesome for the participant resulting in either 1) use of systemic corticosteroids or increase of a stable systemic maintenance dose for a duration of at least 3 consecutive days as prescribed; or 2) participant initiation of systemic corticosteroids for a duration of at least 3 consecutive days. It was considered resolved 7 days after the last dose of OCS administered (10 days after an injectable corticosteroid). Courses of corticosteroids initiated after this time period were considered a separate new asthma exacerbation. Severe AER was evaluated by subgroup FEV1 reversibility. Data were summarized together for 'Placebo, Q2W' and 'Placebo, Q2/4W' arms.
Time Frame: Week 1 up to Week 53
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: AER events/person-year
Arm/Group | Placebo Total | Tralokinumab 300 mg, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Number analyzed (Participants) | 151 | 150 | 151
AER events/person-year
  Reversibility >=12% (n=57,43,49) | 0.11 [0.04 to 0.25] | 0.13 [0.04 to 0.29] | 0.13 [0.05 to 0.28]
  Reversibility <12% (n=91,101,97) | 0.20 [0.12 to 0.32] | 0.10 [0.05 to 0.19] | 0.09 [0.04 to 0.18]
Statistical Analysis 1: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline FEV1 reversibility >=12%; Test type: Superiority or Other; p = 0.975, Poisson regression; Rate Ratio = 1.03, 95% CI 2-sided [0.14 to 7.67] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 2: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline FEV1 reversibility >=12%; Test type: Superiority or Other; p = 0.473, Poisson regression; Rate Ratio = 1.66, 95% CI 2-sided [0.41 to 6.67] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 3: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline FEV1 reversibility <12%; Test type: Superiority or Other; p = 0.099, Poisson regression; Rate Ratio = 0.49, 95% CI 2-sided [0.21 to 1.14] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 4: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline FEV1 reversibility <12%; Test type: Superiority or Other; p = 0.148, Poisson regression; Rate Ratio = 0.42, 95% CI 2-sided [0.13 to 1.36] — [estimate comment as in outcome 21, analysis 1]

29. Secondary Outcome: Severe Asthma Exacerbation Rate (AER) by T-helper-2 (Th2) Status
Description: Severe AER was assessed based on AER data up to Week 53. An asthma exacerbation is a progressive increase of asthma symptoms that does not resolve after the initiation of rescue medications and remains troublesome for the participant resulting in either 1) use of systemic corticosteroids or increase of a stable systemic maintenance dose for a duration of at least 3 days as prescribed; or 2) participant initiation of systemic corticosteroids for a duration of at least 3 days. It was considered resolved 7 days after last dose of OCS administered (10 days after injectable corticosteroid). Courses of corticosteroids initiated after this time period were considered a separate new asthma exacerbation. Severe AER was evaluated by subgroup Th2 status. Th2-high include participants who had IgE >100 IU/mL and blood eosinophils >=0.14*10^9/Liter. Th2 low would include participants who do not meet Th2 high status. Data were summarized together for 'Placebo, Q2W' and 'Placebo, Q2/4W' arms.
Time Frame: Week 1 up to Week 53
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: AER events/person-year
Arm/Group | Placebo Total | Tralokinumab 300 mg, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Number analyzed (Participants) | 151 | 150 | 151
AER events/person-year
  Th2 high (n=70,74,67) | 0.12 [0.05 to 0.24] | 0.12 [0.05 to 0.23] | 0.06 [0.02 to 0.16]
  Th2 Low (n=73,61,72) | 0.21 [0.11 to 0.35] | 0.05 [0.01 to 0.15] | 0.12 [0.05 to 0.24]
Statistical Analysis 1: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Th2 high; Test type: Superiority or Other; p = 0.698, Poisson regression; Rate Ratio = 0.82, 95% CI 2-sided [0.31 to 2.19] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 2: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Th2 high; Test type: Superiority or Other; p = 0.299, Poisson regression; Rate Ratio = 0.55, 95% CI 2-sided [0.18 to 1.70] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 3: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Th2 Low; Test type: Superiority or Other; p = 0.105, Poisson regression; Rate Ratio = 0.25, 95% CI 2-sided [0.05 to 1.34] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 4: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Th2 Low; Test type: Superiority or Other; p = 0.576, Poisson regression; Rate Ratio = 0.70, 95% CI 2-sided [0.20 to 2.47] — [estimate comment as in outcome 21, analysis 1]

30. Secondary Outcome: Severe Asthma Exacerbation Rate (AER) by Baseline Peripheral Blood Eosinophil Count
Description: Severe AER was assessed based on AER data up to Week 53. Annualized AER was assessed based on AER data up to Week 53. An asthma exacerbation defined as a progressive increase of asthma symptoms that does not resolve after the initiation of rescue medications and remains troublesome for the participant resulting in either 1) use of systemic corticosteroids or increase of a stable systemic maintenance dose for a duration of at least 3 consecutive days as prescribed; or 2) participant initiation of systemic corticosteroids for a duration of at least 3 consecutive days. It was considered resolved 7 days after the last dose of OCS administered (10 days after an injectable corticosteroid). Courses of corticosteroids initiated after this time period were considered a separate new asthma exacerbation. Severe AER was evaluated by subgroup baseline peripheral blood eosinophil count. Data were summarized together for 'Placebo, Q2W' and 'Placebo, Q2/4W' arms.
Time Frame: Week 1 up to Week 53
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: AER events/person-year
Arm/Group | Placebo Total | Tralokinumab 300 mg, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Number analyzed (Participants) | 151 | 150 | 151
AER events/person-year
  >= 300 cells/mcgL (n=54,60,50) | 0.22 [0.11 to 0.40] | 0.16 [0.07 to 0.31] | 0.15 [0.06 to 0.31]
  < 300 cells/mcgL (n=89,82,94) | 0.13 [0.07 to 0.24] | 0.08 [0.03 to 0.16] | 0.08 [0.03 to 0.17]
Statistical Analysis 1: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline eosinophil count >=300 cells/mcgL; Test type: Superiority or Other; p = 0.133, Poisson regression; Rate Ratio = 0.48, 95% CI 2-sided [0.19 to 1.25] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 2: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline eosinophil count >=300 cells/mcgL; Test type: Superiority or Other; p = 0.241, Poisson regression; Rate Ratio = 0.46, 95% CI 2-sided [0.13 to 1.67] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 3: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline eosinophil count <300 cells/mcgL; Test type: Superiority or Other; p = 0.510, Poisson regression; Rate Ratio = 0.59, 95% CI 2-sided [0.12 to 2.84] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 4: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline eosinophil count <300 cells/mcgL; Test type: Superiority or Other; p = 0.661, Poisson regression; Rate Ratio = 0.74, 95% CI 2-sided [0.19 to 2.85] — [estimate comment as in outcome 21, analysis 1]

31. Secondary Outcome: Percent Change From Baseline in Prebronchodilator FEV1 at Week 53 in Subgroups
Description: Prebronchodilator FEV1 was evaluated by subgroups. Data were summarized together for 'Placebo, Q2W' and 'Placebo, Q2/4W' arms.
Time Frame: Week 1 up to Week 53
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Placebo Total | Tralokinumab 300 mg, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Number analyzed (Participants) | 151 | 150 | 151
Percent change
  Baseline SP >=median (n=54,71,65) | 4.17 (2.75) [0.88 to 1.43] | 10.48 (3.01) [0.65 to 1.08] | 4.36 (2.25) [1.03 to 1.55]
  Baseline SP <median (n=71,59,56) | 1.23 (2.82) [0.55 to 0.95] | 7.46 (3.00) [0.76 to 1.25] | 1.30 (2.12) [0.45 to 0.85]
  Baseline SP >=25th Percentile (n=88,102,100) | 4.10 (2.29) [0.75 to 1.15] | 10.40 (2.43) [0.67 to 1.03] | 2.31 (1.66) [0.87 to 1.25]
  Baseline SP <25th Percentile (n=37,28,21) | -1.29 (3.92) [0.58 to 1.16] | 4.40 (4.39) [0.81 to 1.56] | 5.99 (4.22) [0.38 to 1.05]
  Baseline SP >=75th Percentile (n=25,40,32) | 2.32 (4.07) [0.76 to 1.60] | 11.05 (4.67) [0.65 to 1.25] | 2.97 (3.33) [1.60 to 2.55]
  Baseline SP <75th Percentile (n=100,90,89) | 2.55 (2.28) [0.69 to 1.04] | 8.25 (2.29) [0.73 to 1.11] | 2.94 (1.75) [0.46 to 0.77]
  Th2 high (n=63,62,57) | 2.10 (2.62) | 11.62 (3.23) | 4.52 (2.39)
  Th2 low (n=57,55,55) | 1.90 (3.09) | 3.87 (2.50) | 0.13 (1.72)
  Baseline PBEC >=150 cells/mcgL (n=81,89,75) | 1.98 (2.32) | 10.97 (2.71) | 4.67 (2.17)
  Baseline PBEC <150 cells/mcgL (n=39,34,40) | 2.05 (3.89) | 5.75 (3.75) | -0.40 (2.00)
  Baseline PBEC >=300 cells/mcgL (n=45,51,39) | 0.59 (2.88) | 14.04 (3.88) | 4.65 (2.90)
  Baseline PBEC <300 cells/mcgL (n=75,72,76) | 2.85 (2.71) | 6.33 (2.57) | 2.01 (1.89)
  Baseline FEV1 reversibility >=12% (n=49,36,41) | 11.02 (3.85) | 22.78 (5.20) | 11.80 (3.48)
  Baseline FEV1 reversibility <12% (n=76,92,80) | -2.99 (1.90) | 3.98 (1.97) | -1.66 (1.28)
  2 asthma exacerbations (n=84,81,82) | 0.76 (2.16) | 8.99 (2.41) | 3.57 (2.04)
  > 2 but < 6 asthma exacerbations (n=41,49,40) | 6.08 (4.12) | 9.32 (4.05) | 1.63 (2.17)
  Chronic OCS use (n=20,21,16) | 3.44 (5.82) | 6.96 (6.56) | -0.48 (5.31)
  Without chronic OCS use (n=105,109,106) | 2.32 (2.10) | 9.52 (2.22) | 3.45 (1.59)
Statistical Analysis 1: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline serum periostin >= median; Test type: Superiority or Other; p = 0.057, Repeated measure model; Difference of LS-mean = 6.79, 95% CI 2-sided [-0.21 to 13.79]
Statistical Analysis 2: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline serum periostin >= median; Test type: Superiority or Other; p = 0.874, Repeated measure model; Difference of LS-mean = 0.57, 95% CI 2-sided [-6.54 to 7.68]
Statistical Analysis 3: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline serum periostin < median; Test type: Superiority or Other; p = 0.028, Repeated measure model; Difference of LS-mean = 7.37, 95% CI 2-sided [0.80 to 13.95]
Statistical Analysis 4: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline serum periostin < median; Test type: Superiority or Other; p = 0.745, Repeated measure model; Difference of LS-mean = 1.09, 95% CI 2-sided [-5.48 to 7.66]
Statistical Analysis 5: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline serum periostin >= 25th percentile; Test type: Superiority or Other; p = 0.011, Repeated measure model; Difference of LS-mean = 7.12, 95% CI 2-sided [1.66 to 12.58]
Statistical Analysis 6: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline serum periostin >= 25th percentile; Test type: Superiority or Other; p = 0.863, Repeated measure model; Difference of LS-mean = -0.48, 95% CI 2-sided [-5.93 to 4.97]
Statistical Analysis 7: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline serum periostin < 25th percentile; Test type: Superiority or Other; p = 0.221, Repeated measure model; Difference of LS-mean = 6.24, 95% CI 2-sided [-3.80 to 16.27]
Statistical Analysis 8: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline serum periostin < 25th percentile; Test type: Superiority or Other; p = 0.108, Repeated measure model; Difference of LS-mean = 8.58, 95% CI 2-sided [-1.91 to 19.07]
Statistical Analysis 9: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline serum periostin >= 75th percentile; Test type: Superiority or Other; p = 0.090, Repeated measure model; Difference of LS-mean = 9.89, 95% CI 2-sided [-1.57 to 21.35]
Statistical Analysis 10: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline serum periostin >= 75th percentile; Test type: Superiority or Other; p = 0.908, Repeated measure model; Difference of LS-mean = 0.70, 95% CI 2-sided [-11.19 to 12.59]
Statistical Analysis 11: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline serum periostin < 75th percentile; Test type: Superiority or Other; p = 0.013, Repeated measure model; Difference of LS-mean = 6.52, 95% CI 2-sided [1.41 to 11.64]
Statistical Analysis 12: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline serum periostin < 75th percentile; Test type: Superiority or Other; p = 0.635, Repeated measure model; Difference of LS-mean = 1.23, 95% CI 2-sided [-3.84 to 6.29]
Statistical Analysis 13: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Th2 high; Test type: Superiority or Other; p = 0.014, Repeated measure model; Difference of LS-mean = 8.89, 95% CI 2-sided [1.84 to 15.94]
Statistical Analysis 14: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Th2 high; Test type: Superiority or Other; p = 0.280, Repeated measure model; Difference of LS-mean = 3.91, 95% CI 2-sided [-3.19 to 11.02]
Statistical Analysis 15: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Th2 low; Test type: Superiority or Other; p = 0.292, Repeated measure model; Difference of LS-mean = 3.22, 95% CI 2-sided [-2.78 to 9.22]
Statistical Analysis 16: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Th2 low; Test type: Superiority or Other; p = 0.691, Repeated measure model; Difference of LS-mean = -1.18, 95% CI 2-sided [-6.99 to 4.64]
Statistical Analysis 17: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline peripheral blood eosinophil count >= 150 cells/μL; Test type: Superiority or Other; p = 0.004, Repeated measure model; Difference of LS-mean = 8.83, 95% CI 2-sided [2.85 to 14.81]
Statistical Analysis 18: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline peripheral blood eosinophil count >= 150 cells/μL; Test type: Superiority or Other; p = 0.177, Repeated measure model; Difference of LS-mean = 4.25, 95% CI 2-sided [-1.92 to 10.43]
Statistical Analysis 19: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline peripheral blood eosinophil count < 150 cells/μL; Test type: Superiority or Other; p = 0.159, Repeated measure model; Difference of LS-mean = 6.05, 95% CI 2-sided [-2.39 to 14.50]
Statistical Analysis 20: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline peripheral blood eosinophil count < 150 cells/μL; Test type: Superiority or Other; p = 0.857, Repeated measure model; Difference of LS-mean = -0.72, 95% CI 2-sided [-8.63 to 7.18]
Statistical Analysis 21: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline peripheral blood eosinophil count >= 300 cells/μL; Test type: Superiority or Other; p = 0.002, Repeated measure model; Difference of LS-mean = 13.75, 95% CI 2-sided [5.28 to 22.22]
Statistical Analysis 22: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline peripheral blood eosinophil count >= 300 cells/μL; Test type: Superiority or Other; p = 0.243, Repeated measure model; Difference of LS-mean = 5.23, 95% CI 2-sided [-3.56 to 14.02]
Statistical Analysis 23: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline peripheral blood eosinophil count < 300 cells/μL; Test type: Superiority or Other; p = 0.144, Repeated measure model; Difference of LS-mean = 4.37, 95% CI 2-sided [-1.50 to 10.24]
Statistical Analysis 24: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline peripheral blood eosinophil count < 300 cells/μ; Test type: Superiority or Other; p = 0.804, Baseline peripheral blood eosinophil cou; Difference of LS-mean = 0.72, 95% CI 2-sided [-5.01 to 6.46]
Statistical Analysis 25: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline FEV1 reversibility >= 12%; Test type: Superiority or Other; p = 0.029, Repeated measure model; Difference of LS-mean = 11.19, 95% CI 2-sided [1.15 to 21.23]
Statistical Analysis 26: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline FEV1 reversibility >= 12%; Test type: Superiority or Other; p = 0.887, Repeated measure model; Difference of LS-mean = 0.72, 95% CI 2-sided [-9.19 to 10.62]
Statistical Analysis 27: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline FEV1 reversibility < 12%; Test type: Superiority or Other; p = 0.002, Repeated measure model; Difference of LS-mean = 7.67, 95% CI 2-sided [2.76 to 12.59]
Statistical Analysis 28: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline FEV1 reversibility < 12%; Test type: Superiority or Other; p = 0.268, Repeated measure model; Difference of LS-mean = 2.79, 95% CI 2-sided [-2.15 to 7.74]
Statistical Analysis 29: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; 2 asthma exacerbations in the past year; Test type: Superiority or Other; p = 0.003, Repeated measure model; Difference of LS-mean = 7.82, 95% CI 2-sided [2.64 to 13.01]
Statistical Analysis 30: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; 2 asthma exacerbations in the past year; Test type: Superiority or Other; p = 0.361, Repeated measure model; Difference of LS-mean = 2.42, 95% CI 2-sided [-2.78 to 7.62]
Statistical Analysis 31: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; > 2 but < 6 asthma exacerbations in the past year; Test type: Superiority or Other; p = 0.185, Repeated measure model; Difference of LS-mean = 6.34, 95% CI 2-sided [-3.06 to 15.75]
Statistical Analysis 32: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; > 2 but < 6 asthma exacerbations in the past year; Test type: Superiority or Other; p = 0.986, Repeated measure model; Difference of LS-mean = -0.08, 95% CI 2-sided [-9.50 to 9.34]
Statistical Analysis 33: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Chronic OCS use; Test type: Superiority or Other; p = 0.912, Repeated measure model; Difference of LS-mean = 0.87, 95% CI 2-sided [-14.70 to 16.44]
Statistical Analysis 34: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Chronic OCS use; Test type: Superiority or Other; p = 0.860, Repeated measure model; Difference of LS-mean = -1.46, 95% CI 2-sided [-17.76 to 14.84]
Statistical Analysis 35: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Without chronic OCS use; Test type: Superiority or Other; p = 0.002, Repeated measure model; Difference of LS-mean = 7.56, 95% CI 2-sided [2.76 to 12.36]
Statistical Analysis 36: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Without chronic OCS use; Test type: Superiority or Other; p = 0.601, Repeated measure model; Difference of LS-mean = 1.28, 95% CI 2-sided [-3.51 to 6.06]

32. Secondary Outcome: Change From Baseline in Mean ACQ-6 Scores at Week 53 in Subgroups
Description: as for outcome 9
Time Frame: Week 1 up to Week 53
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Total | Tralokinumab 300 mg, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Number analyzed (Participants) | 151 | 150 | 151
units on a scale
  Baseline SP >= Median (n= 51, 65, 60) | -0.88 (0.15) [0.88 to 1.43] | -1.18 (0.13) [0.65 to 1.08] | -0.85 (0.14) [1.03 to 1.55]
  Baseline SP < Median (n= 67, 50, 52) | -0.77 (0.14) [0.55 to 0.95] | -0.81 (0.15) [0.76 to 1.25] | -1.03 (0.17) [0.45 to 0.85]
  Baseline SP >= 25th Percentile (n= 82, 92, 91) | -0.86 (0.12) [0.75 to 1.15] | -1.04 (0.11) [0.67 to 1.03] | -0.93 (0.13) [0.87 to 1.25]
  Baseline SP < 25th Percentile (n= 36, 23, 21) | -0.73 (0.19) [0.58 to 1.16] | -0.95 (0.24) [0.81 to 1.56] | -0.92 (0.24) [0.38 to 1.05]
  Baseline SP >= 75th Percentile (n= 25, 34, 27) | -0.75 (0.14) [0.76 to 1.60] | -1.25 (0.18) [0.65 to 1.25] | -1.01 (0.23) [1.60 to 2.55]
  Baseline SP < 75th Percentile (n= 93, 81, 85) | -0.84 (0.12) [0.69 to 1.04] | -0.92 (0.12) [0.73 to 1.11] | -0.91 (0.13) [0.46 to 0.77]
  Th2 High (n= 59, 56, 55) | -0.95 (0.13) | -1.10 (0.15) | -1.02 (0.15)
  Th2 Low (n= 55, 47, 50) | -0.70 (0.16) | -0.94 (0.14) | -0.87 (0.17)
  Baseline EC >= 150 Cells/UL (n= 77, 78, 70) | -0.84 (0.13) | -1.07 (0.13) | -0.94 (0.13)
  Baseline EC < 150 Cells/UL (n= 37, 31, 37) | -0.81 (0.18) | -0.92 (0.16) | -1.02 (0.21)
  Baseline EC >= 300 Cells/UL (n= 43, 44, 37) | -0.77 (0.15) | -1.24 (0.16) | -0.91 (0.17)
  Baseline EC < 300 Cells/UL (n= 71, 65, 70) | -0.86 (0.14) | -0.88 (0.12) | -1.00 (0.15)
  Baseline FEV1 Reversibility >= 12% (n= 43, 33, 35) | -0.47 (0.19) | -0.90 (0.18) | -0.76 (0.20)
  Baseline FEV1 Reversibility < 12% (n= 73, 78, 75) | -1.03 (0.11) | -1.12 (0.12) | -1.02 (0.13)
  2 Asthma Exacerbations (n= 79, 72, 75) | -0.77 (0.13) | -0.94 (0.13) | -0.95 (0.14)
  >2 Asthma Exacerbations (n= 39, 43, 37) | -0.93 (0.17) | -1.15 (0.15) | -0.90 (0.19)
  With Chronic OCS Use (n= 20, 17, 18) | -0.39 (0.25) | -0.89 (0.28) | -0.16 (0.23)
  Without Chronic OCS Use (n= 98, 98, 94) | -0.91 (0.11) | -1.04 (0.11) | -1.08 (0.12)
Statistical Analysis 1: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline serum periostin >= median; Test type: Superiority or Other; p = 0.145, Repeated measure model; Difference of LS-mean = -0.24, 95% CI 2-sided [-0.57 to 0.08]
Statistical Analysis 2: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline serum periostin >= median; Test type: Superiority or Other; p = 0.759, Repeated measure model; Difference of LS-mean = 0.05, 95% CI 2-sided [-0.28 to 0.38]
Statistical Analysis 3: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline serum periostin < median; Test type: Superiority or Other; p = 0.936, Repeated measure model; Difference of LS-mean = -0.01, 95% CI 2-sided [-0.38 to 0.35]
Statistical Analysis 4: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline serum periostin < median; Test type: Superiority or Other; p = 0.127, Repeated measure model; Difference of LS-mean = -0.28, 95% CI 2-sided [-0.64 to 0.08]
Statistical Analysis 5: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline serum periostin>= 25th percentile; Test type: Superiority or Other; p = 0.343, Repeated measure model; Difference of LS-mean = -0.13, 95% CI 2-sided [-0.41 to 0.14]
Statistical Analysis 6: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline serum periostin>= 25th percentile; Test type: Superiority or Other; p = 0.928, Repeated measure model; Difference of LS-mean = -0.01, 95% CI 2-sided [-0.29 to 0.27]
Statistical Analysis 7: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline serum periostin < 25th percentile; Test type: Superiority or Other; p = 0.374, Repeated measure model; Difference of LS-mean = -0.23, 95% CI 2-sided [-0.74 to 0.28]
Statistical Analysis 8: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline serum periostin < 25th percentile; Test type: Superiority or Other; p = 0.259, Repeated measure model; Difference of LS-mean = -0.29, 95% CI 2-sided [-0.81 to 0.22]
Statistical Analysis 9: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline serum periostin >= 75th percentile; Test type: Superiority or Other; p = 0.127, Repeated measure model; Difference of LS-mean = -0.37, 95% CI 2-sided [-0.84 to 0.11]
Statistical Analysis 10: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline serum periostin >= 75th percentile; Test type: Superiority or Other; p = 0.775, Repeated measure model; Difference of LS-mean = -0.07, 95% CI 2-sided [-0.56 to 0.42]
Statistical Analysis 11: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline serum periostin < 75th percentile; Test type: Superiority or Other; p = 0.512, Repeated measure model; Difference of LS-mean = -0.10, 95% CI 2-sided [-0.38 to 0.19]
Statistical Analysis 12: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline serum periostin < 75th percentile; Test type: Superiority or Other; p = 0.404, Repeated measure model; Difference of LS-mean = -0.12, 95% CI 2-sided [-0.40 to 0.16]
Statistical Analysis 13: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Th2 high; Test type: Superiority or Other; p = 0.181, Repeated measure model; Difference of LS-mean = -0.24, 95% CI 2-sided [-0.59 to 0.11]
Statistical Analysis 14: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Th2 high; Test type: Superiority or Other; p = 0.161, Repeated measure model; Difference of LS-mean = -0.25, 95% CI 2-sided [-0.60 to 0.10]
Statistical Analysis 15: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Th2 low; Test type: Superiority or Other; p = 0.540, Repeated measure model; Difference of LS-mean = -0.11, 95% CI 2-sided [-0.47 to 0.25]
Statistical Analysis 16: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Th2 low; Test type: Superiority or Other; p = 0.674, Repeated measure model; Difference of LS-mean = -0.07, 95% CI 2-sided [-0.42 to 0.27]
Statistical Analysis 17: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline peripheral blood eosinophil count >= 150 cells/μL; Test type: Superiority or Other; p = 0.154, Repeated measure model; Difference of LS-mean = -0.22, 95% CI 2-sided [-0.52 to 0.08]
Statistical Analysis 18: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline peripheral blood eosinophil count >= 150 cells/μ; Test type: Superiority or Other; p = 0.271, Repeated measure model; Difference of LS-mean = -0.17, 95% CI 2-sided [-0.48 to 0.13]
Statistical Analysis 19: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline peripheral blood eosinophil count < 150 cells/μL; Test type: Superiority or Other; p = 0.725, Repeated measure model; Difference of LS-mean = -0.08, 95% CI 2-sided [-0.51 to 0.36]
Statistical Analysis 20: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline peripheral blood eosinophil count < 150 cells/μL; Test type: Superiority or Other; p = 0.559, Repeated measure model; Difference of LS-mean = -0.12, 95% CI 2-sided [-0.53 to 0.28]
Statistical Analysis 21: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline peripheral blood eosinophil count >= 300 cells/μL; Test type: Superiority or Other; p = 0.019, Repeated measure model; Difference of LS-mean = -0.47, 95% CI 2-sided [-0.87 to -0.08]
Statistical Analysis 22: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline peripheral blood eosinophil count >= 300 cells/μL; Test type: Superiority or Other; p = 0.348, Repeated measure model; Difference of LS-mean = -0.20, 95% CI 2-sided [-0.61 to 0.21]
Statistical Analysis 23: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline peripheral blood eosinophil count < 300 cells/μL; Test type: Superiority or Other; p = 0.855, Repeated measure model; Difference of LS-mean = -0.03, 95% CI 2-sided [-0.35 to 0.29]
Statistical Analysis 24: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline peripheral blood eosinophil count < 300 cells/μL; Test type: Superiority or Other; p = 0.203, Repeated measure model; Difference of LS-mean = -0.20, 95% CI 2-sided [-0.50 to 0.11]
Statistical Analysis 25: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline FEV1 reversibility >= 12%; Test type: Superiority or Other; p = 0.055, Repeated measure model; Difference of LS-mean = -0.44, 95% CI 2-sided [-0.89 to 0.01]
Statistical Analysis 26: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline FEV1 reversibility >= 12%; Test type: Superiority or Other; p = 0.104, Repeated measure model; Difference of LS-mean = -0.37, 95% CI 2-sided [-0.82 to 0.08]
Statistical Analysis 27: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline FEV1 reversibility < 12%; Test type: Superiority or Other; p = 0.652, Repeated measure model; Difference of LS-mean = -0.07, 95% CI 2-sided [-0.37 to 0.23]
Statistical Analysis 28: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline FEV1 reversibility < 12%; Test type: Superiority or Other; p = 0.905, Repeated measure model; Difference of LS-mean = 0.02, 95% CI 2-sided [-0.28 to 0.32]
Statistical Analysis 29: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; 2 asthma exacerbations in the past year; Test type: Superiority or Other; p = 0.198, Repeated measure model; Difference of LS-mean = -0.19, 95% CI 2-sided [-0.49 to 0.10]
Statistical Analysis 30: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; 2 asthma exacerbations in the past year; Test type: Superiority or Other; p = 0.226, Repeated measure model; Difference of LS-mean = -0.18, 95% CI 2-sided [-0.47 to 0.11]
Statistical Analysis 31: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; > 2 but < 6 asthma exacerbations in the past year; Test type: Superiority or Other; p = 0.513, Repeated measure model; Difference of LS-mean = -0.14, 95% CI 2-sided [-0.56 to 0.28]
Statistical Analysis 32: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; > 2 but < 6 asthma exacerbations in the past year; Test type: Superiority or Other; p = 0.974, Repeated measure model; Difference of LS-mean = -0.01, 95% CI 2-sided [-0.43 to 0.42]
Statistical Analysis 33: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Chronic OCS use; Test type: Superiority or Other; p = 0.226, Repeated measure model; Difference of LS-mean = -0.37, 95% CI 2-sided [-0.97 to 0.23]
Statistical Analysis 34: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Chronic OCS use; Test type: Superiority or Other; p = 0.613, Repeated measure model; Difference of LS-mean = 0.15, 95% CI 2-sided [-0.44 to 0.75]
Statistical Analysis 35: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Without chronic OCS use; Test type: Superiority or Other; p = 0.198, Repeated measure model; Difference of LS-mean = -0.17, 95% CI 2-sided [-0.43 to 0.09]
Statistical Analysis 36: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Without chronic OCS use; Test type: Superiority or Other; p = 0.165, Repeated measure model; Difference of LS-mean = -0.19, 95% CI 2-sided [-0.45 to 0.08]

33. Secondary Outcome: Change From Baseline in Total AQLQ(S) Scores at Week 53 in Subgroups
Description: as for outcome 10
Time Frame: Week 1 up to Week 53
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Total | Tralokinumab 300 mg, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Number analyzed (Participants) | 151 | 150 | 151
units on a scale
  Baseline SP >= Median (n= 46, 63, 56) | 0.89 (0.15) [0.88 to 1.43] | 1.10 (0.14) [0.65 to 1.08] | 0.95 (0.17) [1.03 to 1.55]
  Baseline SP < Median ( n= 61, 46, 45) | 0.82 (0.14) [0.55 to 0.95] | 0.95 (0.15) [0.76 to 1.25] | 1.07 (0.17) [0.45 to 0.85]
  Baseline SP >= 25th Percentile (n= 73, 88, 82) | 0.87 (0.12) [0.75 to 1.15] | 1.08 (0.11) [0.67 to 1.03] | 0.98 (0.14) [0.87 to 1.25]
  Baseline SP < 25th Percentile (n= 34, 21, 19) | 0.81 (0.19) [0.58 to 1.16] | 0.84 (0.24) [0.81 to 1.56] | 1.09 (0.24) [0.38 to 1.05]
  Baseline SP >= 75th Percentile (n= 23, 33, 24) | 0.76 (0.17) [0.76 to 1.60] | 1.20 (0.19) [0.65 to 1.25] | 1.13 (0.28) [1.60 to 2.55]
  Baseline SP < 75th Percentile (n= 84, 76, 77) | 0.87 (0.12) [0.69 to 1.04] | 0.97 (0.12) [0.73 to 1.11] | 0.96 (0.13) [0.46 to 0.77]
  Th2 high (n=54,52,50) | 0.88 (0.13) | 1.12 (0.15) | 1.12 (0.18)
  Th2 low (n= 49, 45, 44 ) | 0.79 (0.17) | 0.88 (0.15) | 0.94 (0.17)
  Baseline EC >= 150 Cells/UL (n=69, 72, 64) | 0.91 (0.11) | 1.06 (0.13) | 1.02 (0.15)
  Baseline EC< 150 Cells/UL (n= 34, 31, 32) | 0.68 (0.20) | 0.93 (0.13) | 1.05 (0.20)
  Baseline EC >= 300 Cells/UL (n= 39, 40, 35) | 0.81 (0.15) | 0.98 (0.17) | 0.82 (0.20)
  Baseline EC < 300 Cells/UL (N= 64, 63, 61) | 0.84 (0.14) | 1.05 (0.13) | 1.15 (0.15)
  Baseline FEV1 Reversibility >= 12% (n= 39, 29, 32) | 0.75 (0.17) | 1.14 (0.16) | 0.95 (0.22)
  Baseline FEV1 Reversibility < 12% (n= 66, 76, 67) | 0.94 (0.13) | 1.04 (0.13) | 1.04 (0.14)
  2 Asthma Exacerbations (n=73, 68, 68) | 0.88 (0.13) | 1.09 (0.14) | 1.14 (0.15)
  >2 Asthma Exacerbations (n= 34, 41, 33) | 0.78 (0.16) | 0.96 (0.14) | 0.73 (0.20)
  With Chronic OCS Use (n= 17, 16, 16) | 0.53 (0.19) | 0.87 (0.29) | 0.26 (0.26)
  Without Chronic OCS Use (n= 90, 93, 85) | 0.91 (0.11) | 1.07 (0.11) | 1.14 (0.13)
Statistical Analysis 1: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline serum periostin >= median; Test type: Superiority or Other; p = 0.211, Repeated measure model; Difference of LS-mean = 0.23, 95% CI 2-sided [-0.13 to 0.60]
Statistical Analysis 2: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline serum periostin >= median; Test type: Superiority or Other; p = 0.397, Repeated measure model; Difference of LS-mean = 0.16, 95% CI 2-sided [-0.21 to 0.53]
Statistical Analysis 3: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline serum periostin < median; Test type: Superiority or Other; p = 0.315, Repeated Measure Model; Difference of LS-mean = 0.19, 95% CI 2-sided [-0.18 to 0.56]
Statistical Analysis 4: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline serum periostin < median; Test type: Superiority or Other; p = 0.166, Repeated measure model; Difference of LS-mean = 0.26, 95% CI 2-sided [-0.11 to 0.63]
Statistical Analysis 5: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline serum periostin >= 25th percentile; Test type: Superiority or Other; p = 0.262, Repeated measure model; Difference of LS-mean = 0.17, 95% CI [-0.13 to 0.47]
Statistical Analysis 6: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline serum periostin >= 25th percentile; Test type: Superiority or Other; p = 0.379, Repeated measure model; Difference of LS-mean = 0.14, 95% CI 2-sided [-0.17 to 0.44]
Statistical Analysis 7: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline serum periostin < 25th percentile; Test type: Superiority or Other; p = 0.387, Repeated measure model; Difference of LS-mean = 0.25, 95% CI 2-sided [-0.32 to 0.81]
Statistical Analysis 8: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline serum periostin < 25th percentile; Test type: Superiority or Other; p = 0.303, Repeated measure model; Difference of LS-mean = 0.29, 95% CI 2-sided [-0.26 to 0.84]
Statistical Analysis 9: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline serum periostin >=75th percentile; Test type: Superiority or Other; p = 0.127, Repeated measure model; Difference of LS-mean = -0.37, 95% CI 2-sided [-0.84 to 0.11]
Statistical Analysis 10: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline serum periostin >=75th percentile; Test type: Superiority or Other; p = 0.775, Repeated measure model; Difference of LS-mean = -0.07, 95% CI 2-sided [-0.56 to 0.42]
Statistical Analysis 11: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline serum periostin < 75th percentile; Test type: Superiority or Other; p = 0.512, Repeated measure model; Difference of LS-mean = -0.10, 95% CI 2-sided [-0.38 to 0.19]
Statistical Analysis 12: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline serum periostin < 75th percentile; Test type: Superiority or Other; p = 0.404, Repeated measure model; Difference of LS-mean = -0.12, 95% CI 2-sided [-0.40 to 0.16]
Statistical Analysis 13: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Th2 high; Test type: Superiority or Other; p = 0.102, Repeated measure model; Difference of LS-mean = 0.31, 95% CI 2-sided [-0.06 to 0.69]
Statistical Analysis 14: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Th2 high; Test type: Superiority or Other; p = 0.116, Repeated measure model; Difference of LS-mean = 0.30, 95% CI 2-sided [-0.08 to 0.68]
Statistical Analysis 15: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Th2 low; Test type: Superiority or Other; p = 0.540, Repeated measure model; Difference of LS-mean = -0.11, 95% CI 2-sided [-0.47 to 0.25]
Statistical Analysis 16: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Th2 low; Test type: Superiority or Other; p = 0.674, Repeated measure model; Difference of LS-mean = -0.07, 95% CI 2-sided [-0.42 to 0.27]
Statistical Analysis 17: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline peripheral blood eosinophil count >=150 cells/μL; Test type: Superiority or Other; p = 0.295, Repeated measure model; Difference of LS-mean = 0.17, 95% CI 2-sided [-0.15 to 0.49]
Statistical Analysis 18: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline peripheral blood eosinophil count >=150 cells/μL; Test type: Superiority or Other; p = 0.342, Repeated measure model; Difference of LS-mean = 0.16, 95% CI 2-sided [-0.17 to 0.49]
Statistical Analysis 19: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline peripheral blood eosinophil count < 150 cells/μL; Test type: Superiority or Other; p = 0.406, Repeated measure model; Difference of LS-mean = 0.18, 95% CI 2-sided [-0.24 to 0.60]
Statistical Analysis 20: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline peripheral blood eosinophil count < 150 cells/μL; Test type: Superiority or Other; p = 0.069, Repeated measure model; Difference of LS-mean = 0.38, 95% CI 2-sided [-0.03 to 0.79]
Statistical Analysis 21: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline peripheral blood eosinophil count >= 300 cells/μL; Test type: Superiority or Other; p = 0.371, Repeated measure model; Difference of LS-mean = 0.19, 95% CI 2-sided [-0.23 to 0.62]
Statistical Analysis 22: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline peripheral blood eosinophil count >= 300 cells/μL; Test type: Superiority or Other; p = 0.766, Repeated measure model; Difference of LS-mean = 0.07, 95% CI 2-sided [-0.37 to 0.51]
Statistical Analysis 23: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline peripheral blood eosinophil count < 300 cells/μL; Test type: Superiority or Other; p = 0.147, Repeated measure model; Difference of LS-mean = 0.24, 95% CI 2-sided [-0.09 to 0.57]
Statistical Analysis 24: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline peripheral blood eosinophil count < 300 cells/μL; Test type: Superiority or Other; p = 0.031, Repeated measure model; Difference of LS-mean = 0.35, 95% CI 2-sided [0.03 to 0.68]
Statistical Analysis 25: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline FEV1 reversibility >= 12%; Test type: Superiority or Other; p = 0.020, Repeated measure model; Difference of LS-mean = 0.59, 95% CI 2-sided [0.10 to 1.09]
Statistical Analysis 26: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline FEV1 reversibility >= 12%; Test type: Superiority or Other; p = 0.226, Repeated measure model; Difference of LS-mean = 0.29, 95% CI 2-sided [-0.18 to 0.77]
Statistical Analysis 27: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Baseline FEV1 reversibility < 12%; Test type: Superiority or Other; p = 0.964, Repeated measure model; Difference of LS-mean = 0.01, 95% CI 2-sided [-0.31 to 0.33]
Statistical Analysis 28: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Baseline FEV1 reversibility < 12%; Test type: Superiority or Other; p = 0.533, Repeated measure model; Difference of LS-mean = 0.10, 95% CI 2-sided [-0.22 to 0.42]
Statistical Analysis 29: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; 2 asthma exacerbations in the past year; Test type: Superiority or Other; p = 0.292, Repeated measure model; Difference of LS-mean = 0.17, 95% CI 2-sided [-0.15 to 0.50]
Statistical Analysis 30: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; 2 asthma exacerbations in the past year; Test type: Superiority or Other; p = 0.097, Repeated measure model; Difference of LS-mean = 0.27, 95% CI 2-sided [-0.05 to 0.59]
Statistical Analysis 31: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; > 2 but < 6 asthma exacerbations in the past year; Test type: Superiority or Other; p = 0.260, Repeated measure model; Difference of LS-mean = 0.24, 95% CI 2-sided [-0.18 to 0.67]
Statistical Analysis 32: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; > 2 but < 6 asthma exacerbations in the past year; Test type: Superiority or Other; p = 0.648, Repeated measure model; Difference of LS-mean = 0.10, 95% CI 2-sided [-0.33 to 0.53]
Statistical Analysis 33: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Chronic OCS use; Test type: Superiority or Other; p = 0.398, Repeated measure model; Difference of LS-mean = 0.28, 95% CI 2-sided [-0.37 to 0.93]
Statistical Analysis 34: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Chronic OCS use; Test type: Superiority or Other; p = 0.327, Repeated measure model; Difference of LS-mean = -0.32, 95% CI 2-sided [-0.95 to 0.32]
Statistical Analysis 35: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Without chronic OCS use; Test type: Superiority or Other; p = 0.105, Repeated measure model; Difference of LS-mean = 0.23, 95% CI 2-sided [-0.05 to 0.52]
Statistical Analysis 36: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Without chronic OCS use; Test type: Superiority or Other; p = 0.030, Repeated measure model; Difference of LS-mean = 0.31, 95% CI 2-sided [0.03 to 0.60]

34. Secondary Outcome: Annual Asthma Exacerbation Rate (AER) by Atopic Asthma Status
Description: Annualized AER was assessed based on AER data up to Week 53. An asthma exacerbation defined as a progressive increase of asthma symptoms that does not resolve after the initiation of rescue medications and remains troublesome for the participant resulting in either 1) use of systemic corticosteroids or increase of a stable systemic maintenance dose for a duration of at least 3 consecutive days as prescribed; or 2) participant initiation of systemic corticosteroids for a duration of at least 3 consecutive days. AER was evaluated by subgroup Atopic and Non-atopic asthma status. Data were summarized together for 'Placebo, Q2W' and 'Placebo, Q2/4W' arms.
Time Frame: Week 1 up to Week 53
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: AER events/person-year
Arm/Group | Placebo Total | Tralokinumab 300 mg, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Number analyzed (Participants) | 151 | 150 | 151
AER events/person-year
  Atopic asthma (n=96,105,92) | 0.85 [0.67 to 1.06] | 0.90 [0.73 to 1.11] | 0.85 [0.67 to 1.06]
  Non-atopic asthma (n=51,42,55) | 1.05 [0.77 to 1.39] | 0.82 [0.56 to 1.15] | 1.10 [0.82 to 1.44]
Statistical Analysis 1: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Atopic asthma; Test type: Superiority or Other; p = 0.803, Poisson regression; Rate Ratio = 0.95, 95% CI 2-sided [0.62 to 1.44] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 2: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Atopic asthma; Test type: Superiority or Other; p = 0.457, Poisson regression; Rate Ratio = 0.83, 95% CI 2-sided [0.52 to 1.35] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 3: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Non-atopic asthma; Test type: Superiority or Other; p = 0.250, Poisson regression; Rate Ratio = 0.71, 95% CI 2-sided [0.40 to 1.27] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 4: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Non-atopic asthma; Test type: Superiority or Other; p = 0.794, Poisson regression; Rate Ratio = 1.07, 95% CI 2-sided [0.66 to 1.74] — [estimate comment as in outcome 21, analysis 1]

35. Secondary Outcome: Annual Asthma Exacerbation Rate (AER) by Chronic OCS Use
Description: Annualized AER was assessed based on AER data up to Week 53. An asthma exacerbation defined as a progressive increase of asthma symptoms that does not resolve after the initiation of rescue medications and remains troublesome for the participant resulting in either 1) use of systemic corticosteroids or increase of a stable systemic maintenance dose for a duration of at least 3 consecutive days as prescribed; or 2) participant initiation of systemic corticosteroids for a duration of at least 3 consecutive days. It was considered resolved 7 days after the last dose of OCS administered (10 days after an injectable corticosteroid). Courses of corticosteroids initiated after this time period were considered a separate new asthma exacerbation. AER evaluated by subgroup chronic OCS use. Data were summarized together for 'Placebo, Q2W' and 'Placebo, Q2/4W' arms.
Time Frame: Week 1 up to Week 53
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: AER events/person-year
Arm/Group | Placebo Total | Tralokinumab 300 mg, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Number analyzed (Participants) | 151 | 150 | 151
AER events/person-year
  With chronic OCS use (n=27,26,24) | 1.37 [0.93 to 1.94] | 2.04 [1.51 to 2.69] | 2.2 [1.62 to 2.91]
  Without chronic OCS use (124,124,127) | 0.81 [0.66 to 1.00] | 0.68 [0.54 to 0.84] | 0.74 [0.59 to 0.91]
Statistical Analysis 1: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; With chronic OCS use; Test type: Superiority or Other; p = 0.614, Poisson regression; Rate Ratio = 1.20, 95% CI 2-sided [0.59 to 2.46] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 2: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; With chronic OCS use; Test type: Superiority or Other; p = 0.506, Poisson regression; Rate Ratio = 1.29, 95% CI 2-sided [0.61 to 2.74] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 3: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2W - Cohort 1; Without chronic OCS use; Test type: Superiority or Other; p = 0.243, Poisson regression; Rate Ratio = 0.79, 95% CI [0.53 to 1.18] — [estimate comment as in outcome 21, analysis 1]
Statistical Analysis 4: Comparison: Placebo Total vs Tralokinumab 300 mg, Q2/4W - Cohort 2; Without chronic OCS use; Test type: Superiority or Other; p = 0.531, Poisson regression; Rate Ratio = 0.87, 95% CI 2-sided [0.57 to 1.34] — [estimate comment as in outcome 21, analysis 1]

36. Secondary Outcome: Change From Baseline in Percentage of Nighttime Awakening at Week 53
Description: Scores for nighttime awakenings were generated based on the single item (question 5) that had a dichotomous response option (YES/NO). Nighttime awakenings were averaged weekly for participants with at least 4 non-missing records each week. The baseline score was calculated with data from Day -7 to Day -1. Data were summarized together for 'Placebo, Q2W' and 'Placebo, Q2/4W' arms.
Time Frame: Day -7 - Day -1 (Baseline) and Day 365 - Day 371 (Week 53)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Placebo Total | Tralokinumab 300 mg, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Number analyzed (Participants) | 151 | 150 | 151
percentage change
  Day -7 - Day -1 (Baseline) (n=151,147,145) | 0.44 (0.42) | 0.42 (0.43) | 0.43 (0.43)
  Change at Day 365 - Day 371 (n=113,108,108) | -0.22 (0.43) | -0.18 (0.37) | -0.23 (0.45)

37. Secondary Outcome: Change From Baseline in Overall Activity Limitations at Week 53
Description: There were 3 activity limitation questions in the ASMA diary. All activity questions were scored from 0 to 4 and averaged, where the higher score indicated greater limitation. Activity limitation scores were averaged weekly for participants with at least 4 non-missing records each week. The baseline score was calculated from Day -7 to Day -1. Data were summarized together for 'Placebo, Q2W' and 'Placebo, Q2/4W' arms.
Time Frame: Day -7 - Day -1 (Baseline) and Day 365 - Day 371 (Week 53)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Total | Tralokinumab 300 mg, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Number analyzed (Participants) | 151 | 150 | 151
units on a scale
  Day -7 - Day -1 (Baseline) (n=151,147,145) | 1.71 (0.86) | 1.52 (0.90) | 1.63 (0.85)
  Change at Day 365 - Day 371 (n=113,108,108) | -0.45 (0.81) | -0.38 (0.84) | -0.48 (0.87)

38. Secondary Outcome: Percent Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) at Week 53
Description: Pre- and post-bronchodilator FEV1 at clinic visits (morning) were measured. FEV1 was the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration. Data were summarized together for 'Placebo, Q2W' and 'Placebo, Q2/4W' arms. Baseline for FEV1 was measured in liters.
Time Frame: Baseline and Week 53
Population: as for outcome 2
Measure: Mean (Standard Error); unit: percentage change in liters
Arm/Group | Placebo Total | Tralokinumab 300 mg, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Number analyzed (Participants) | 151 | 150 | 151
percentage change in liters
  Pre-bronchodilator(BD): Baseline (n=147,146,146) | 1.926 (0.050) | 1.922 (0.056) | 1.934 (0.059)
  Post-BD: Baseline (n=147,141,146) | 2.153 (0.053) | 2.094 (0.061) | 2.110 (0.061)
  Pre-BD:Change from baseline to W53 (n=125,130,122) | 2.50 (1.99) | 9.11 (2.13) | 2.94 (1.54)
  Post-BD:Change from baseline to W53(n=125,126,120) | -1.65 (1.39) | 5.98 (1.85) | 0.18 (1.25)

39. Secondary Outcome: Percent Change From Baseline in Forced Expiratory Volume in 6 Second (FEV6) at Week 53
Description: Pre- and post-bronchodilator FEV6 at clinic visits (morning) were measured. FEV6 was the maximal volume of air exhaled in the six second of a forced expiration from a position of full inspiration. Data were summarized together for 'Placebo, Q2W' and 'Placebo, Q2/4W' arms. Baseline for FEV6 was measured in liters.
Time Frame: Baseline and Week 53
Population: as for outcome 2
Measure: Mean (Standard Error); unit: percentage change in liters
Arm/Group | Placebo Total | Tralokinumab 300 mg, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Number analyzed (Participants) | 151 | 150 | 151
percentage change in liters
  Pre-bronchodilator(BD): Baseline (n=147,146,146) | 2.830 (0.064) | 2.809 (0.072) | 2.827 (0.074)
  Post-BD: Baseline (n=147,141,146) | 3.055 (0.067) | 2.981 (0.075) | 2.980 (0.076)
  Pre-BD:Change from baseline to W53 (n=125,130,122) | 1.06 (1.29) | 5.75 (1.53) | 1.10 (1.18)
  Post-BD:Change from baseline to W53(n=125,126,120) | -1.16 (1.04) | 3.27 (1.36) | -0.11 (1.01)

40. Secondary Outcome: Percent Change From Baseline in Forced Vital Capacity (FVC) at Week 53
Description: Pre- and post-bronchodilator FVC at clinic visits (morning) were measured. FVC was the volume of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. Data were summarized together for 'Placebo, Q2W' and 'Placebo, Q2/4W' arms. Baseline for FVC was measured in liters.
Time Frame: Baseline and Week 53
Population: as for outcome 2
Measure: Mean (Standard Error); unit: percentage change in liters
Arm/Group | Placebo Total | Tralokinumab 300 mg, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Number analyzed (Participants) | 151 | 150 | 151
percentage change in liters
  Pre-bronchodilator(BD): Baseline (n=147,146,146) | 3.003 (0.069) | 2.955 (0.075) | 2.993 (0.079)
  Post-BD: Baseline (n=147,141,146) | 3.225 (0.072) | 3.133 (0.078) | 3.125 (0.080)
  Pre-BD:Change from baseline to W53 (n=125,130,122) | 0.87 (1.31) | 5.43 (1.60) | 0.46 (1.17)
  Post-BD:Change from baseline to W53(n=125,126,120) | -1.51 (1.01) | 2.56 (1.27) | -0.26 (1.03)

41. Secondary Outcome: Percent Change From Baseline in Inspiratory Capacity (IC) at Week 53
Description: Pre- and post-bronchodilator IC at clinic visits (morning) were measured. IC was measured by spirometry. Data were summarized together for 'Placebo, Q2W' and 'Placebo, Q2/4W' arms. Baseline for IC was measured in liters.
Time Frame: Baseline and Week 53
Population: as for outcome 2
Measure: Mean (Standard Error); unit: percentage change in liters
Arm/Group | Placebo Total | Tralokinumab 300 mg, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Number analyzed (Participants) | 151 | 150 | 151
percentage change in liters
  Pre-bronchodilator(BD): Baseline (n=140,138,143) | 0.022 (0.001) | 0.023 (0.001) | 0.023 (0.001)
  Post-BD: Baseline (n=140,133,135) | 0.024 (0.001) | 0.024 (0.001) | 0.024 (0.001)
  Pre-BD:Change from baseline to W53 (n=108,109,103) | 8.56 (3.42) | 0.15 (2.21) | 11.38 (3.71)
  Post-BD:Change from baseline to W53(n=108,109,104) | 3.64 (3.17) | 8.33 (3.14) | 3.17 (2.91)

42. Secondary Outcome: Percent Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) at Week 53 at Home
Description: as for outcome 7
Time Frame: Day 1 - Day 7 (Baseline) and Day 365 - Day 371 (Week 53)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | Placebo Total | Tralokinumab 300 mg, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Number analyzed (Participants) | 151 | 150 | 151
percentage change
  Change at Day 365-371: Morning (n=123,119,113) | -4.96 (3.27) | 1.67 (2.83) | 1.70 (5.41)
  Change at Day 365-371: Evening (n=119,116,111) | -2.83 (3.01) | -2.69 (3.17) | -5.78 (3.63)

43. Secondary Outcome: Percent Change From Baseline in Peak Expiratory Flow (PEF) at Week 53 at Home
Description: as for outcome 8
Time Frame: Day 1 - Day 7 (Baseline) and Day 365 - Day 371 (Week 53)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | Placebo Total | Tralokinumab 300 mg, Q2W - Cohort 1 | Tralokinumab 300 mg, Q2/4W - Cohort 2
Number analyzed (Participants) | 151 | 150 | 151
percentage change
  Change at Day 365-371: Morning (n=123,119,113) | -6.89 (3.09) | -0.64 (3.26) | -2.80 (5.41)
  Change at Day 365-371: Evening (n=129,116,111) | -4.95 (2.99) | -6.62 (3.13) | -11.45 (3.33)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 75
Description: The safety population included all subjects who received any investigational product and had safety data available.
Groups:
- Tralokinumab 300 mg Q2W: Participants received tralokinumab 300 milligram (mg) subcutaneous injection every 2 weeks (Q2W) for a total of 26 doses up to 50 weeks.
- Tralokinumab 300 mg Q2/4W: Participants received tralokinumab 300 mg subcutaneous injection every 2 weeks (Q2W) for 12 weeks followed by every 4 weeks (Q4W) for 38 weeks (Q2/4W) for a total of 16 doses.
Arm/Group | Placebo Total | Tralokinumab 300 mg Q2W | Tralokinumab 300 mg Q2/4W
Serious Adverse Events (participants affected / at risk) | 21/151 | 18/150 | 25/151
Other Adverse Events (participants affected / at risk) | 128/151 | 133/150 | 128/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Total (N=151) | Tralokinumab 300 mg Q2W (N=150) | Tralokinumab 300 mg Q2/4W (N=151)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 2 (3)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic gastropathy (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Femoral hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Amoebiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Beta haemolytic streptococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 3 (3) | 2 (2)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Accidental poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Testicular injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Menometrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 6 (9) | 9 (13) | 10 (13)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Total (N=151) | Tralokinumab 300 mg Q2W (N=150) | Tralokinumab 300 mg Q2/4W (N=151)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 5 (5) | 3 (3)
Conjunctivitis allergic (Eye disorders) | 2 (2) | 3 (3) | 2 (2)
Eye pruritus (Eye disorders) | 0 (0) | 2 (2) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 9 (12) | 1 (1) | 1 (3)
Abdominal pain upper (Gastrointestinal disorders) | 3 (4) | 1 (4) | 2 (2)
Constipation (Gastrointestinal disorders) | 4 (5) | 3 (3) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 12 (19) | 5 (7) | 7 (10)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 4 (5) | 1 (1) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 (6) | 4 (4) | 2 (2)
Nausea (Gastrointestinal disorders) | 7 (15) | 2 (7) | 3 (4)
Toothache (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 8 (20) | 4 (6) | 1 (2)
Administration site rash (General disorders) | 0 (0) | 3 (13) | 3 (3)
Asthenia (General disorders) | 6 (8) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (3) | 2 (4) | 3 (4)
Injection site erythema (General disorders) | 1 (1) | 12 (58) | 7 (15)
Injection site haemorrhage (General disorders) | 3 (3) | 1 (3) | 2 (3)
Injection site pain (General disorders) | 15 (90) | 7 (23) | 11 (61)
Injection site pruritus (General disorders) | 1 (1) | 8 (12) | 1 (2)
Injection site reaction (General disorders) | 0 (0) | 7 (32) | 2 (4)
Injection site swelling (General disorders) | 2 (3) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 6 (10) | 2 (3) | 4 (6)
Acute sinusitis (Infections and infestations) | 5 (6) | 2 (2) | 3 (4)
Bronchitis (Infections and infestations) | 22 (48) | 27 (44) | 20 (27)
Cystitis (Infections and infestations) | 4 (4) | 2 (2) | 1 (1)
Gastroenteritis (Infections and infestations) | 9 (9) | 7 (9) | 6 (6)
Herpes zoster (Infections and infestations) | 3 (3) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 13 (15) | 11 (13) | 14 (15)
Lower respiratory tract infection (Infections and infestations) | 4 (5) | 3 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 40 (83) | 35 (57) | 26 (62)
Oral candidiasis (Infections and infestations) | 3 (5) | 6 (6) | 2 (2)
Pharyngitis (Infections and infestations) | 9 (15) | 6 (9) | 11 (18)
Pneumonia (Infections and infestations) | 3 (3) | 2 (2) | 3 (3)
Respiratory tract infection (Infections and infestations) | 3 (4) | 6 (10) | 1 (1)
Rhinitis (Infections and infestations) | 9 (10) | 5 (5) | 8 (9)
Sinusitis (Infections and infestations) | 10 (15) | 5 (5) | 8 (10)
Upper respiratory tract infection (Infections and infestations) | 18 (28) | 20 (36) | 20 (25)
Urinary tract infection (Infections and infestations) | 9 (19) | 11 (16) | 8 (8)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 4 (5)
Contusion (Injury, poisoning and procedural complications) | 2 (8) | 3 (6) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 3 (4) | 1 (3) | 2 (2)
Foot fracture (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | 2 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 5 (6)
Rib fracture (Injury, poisoning and procedural complications) | 1 (2) | 3 (3) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (8) | 10 (15) | 9 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (11) | 8 (11) | 10 (12)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (8) | 6 (6)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (7) | 8 (11)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (6) | 2 (2) | 8 (9)
Dizziness (Nervous system disorders) | 9 (17) | 2 (3) | 3 (3)
Headache (Nervous system disorders) | 17 (36) | 17 (38) | 17 (22)
Migraine (Nervous system disorders) | 3 (14) | 1 (2) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 3 (3) | 6 (6)
Insomnia (Psychiatric disorders) | 4 (4) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 73 (175) | 68 (192) | 58 (188)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (9) | 7 (7) | 8 (11)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 4 (4) | 3 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 7 (16)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 3 (3) | 6 (7)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 1 (1) | 1 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 11 (13) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5) | 1 (1)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 3 (5) | 4 (9)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 1 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (6) | 3 (3) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 7 (7) | 3 (3)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 4 (7) | 3 (3) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 3 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 5 (6) | 2 (2) | 2 (2)
Hypertension (Vascular disorders) | 6 (8) | 8 (8) | 9 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.